CLINICAL TRIAL: NCT00391872
Title: A Randomised, Double-blind, Parallel Group, Phase 3, Efficacy and Safety Study of Ticagrelor Compared With Clopidogrel for Prevention of Vascular Events in Patients With Non-ST or ST Elevation Acute Coronary Syndromes (ACS) [PLATO- a Study of PLATelet Inhibition and Patient Outcomes]
Brief Title: A Comparison of Ticagrelor (AZD6140) and Clopidogrel in Patients With Acute Coronary Syndrome
Acronym: PLATO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D5130C05262; PLATO
Record Dates: First submitted 2006-10-23; First posted 2006-10-25 (Estimated); Results first posted 2012-03-13 (Estimated); Last update posted 2012-03-13 (Estimated); Status verified 2012-02

CONDITIONS: Acute Coronary Syndrome
Keywords: ACS; Acute coronary syndrome; Heart attack; Unstable angina; Coronary artery disease
MeSH Terms: conditions — Acute Coronary Syndrome; Myocardial Infarction; Angina, Unstable; Coronary Artery Disease | interventions — Ticagrelor; Clopidogrel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Clopidogrel (Active Comparator): Oral treatment
  Interventions: Drug: Clopidogrel
- Ticagrelor (Experimental): Oral treatment
  Interventions: Drug: Ticagrelor

INTERVENTIONS:
Drug: Ticagrelor — Ticagrelor (AZD6140) 90 mg twice daily dose (BD)
  Other Names: AZD6140
  Arms: Ticagrelor
Drug: Clopidogrel — Clopidogrel 75 mg once daily dose (ODD)
  Other Names: Plavix®
  Arms: Clopidogrel

SUMMARY:
Ticagrelor is a new, reversible binding, anti-platelet medication. Anti-platelet medications work to prevent the formation of blood clots. Ticagrelor is being developed as a treatment for patients with acute coronary syndrome (ACS). ACS is a term that is used to describe both heart attacks in progress or the imminent threat of a heart attack. ACS is usually caused by the formation of a blood clot in an artery that partially or totally blocks the blood supply to a portion of the heart muscle. Ticagrelor will be compared with clopidogrel to determine which drug, when either is used in conjunction with aspirin, is better at reducing deaths from vascular causes, future heart attacks and/or strokes in patients with ACS.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 18 years or older who has been hospitalised for chest pain and potential ACS
* Females of child-bearing potential must have a negative pregnancy test at enrollment and be willing to use 2 methods of reliable contraception

Exclusion Criteria:

* Persons with moderate or severe liver disease
* Persons who have already been treated with an invasive (angioplasty) procedure for the current episode of ACS
* Persons who are being treated with blood clotting agents that cannot be stopped

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18624 (Actual)
Dates: Start 2006-10; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Harrington, MD, Principal Investigator — Duke Clinical Research Institute; Lars Wallentin, MD, Principal Investigator — Uppsala Clinical Research Centre; Jonathan C. Fox, MD, Study Director — AstraZeneca
Locations (672):
- United States (139):
  - Research Site, Birmingham, Alabama
  - Research Site, Huntsville, Alabama
  - Research Site, Mobile, Alabama
  - Research Site, Tucson, Arizona
  - Research Site, Bakersfield, California
  - Research Site, Beverly Hills, California
  - Research Site, Burbank, California
  - Research Site, Healdsburg, California
  - Research Site, Los Angeles, California
  - Research Site, Roseville, California
  - Research Site, Sacramento, California
  - Research Site, San Diego, California
  - Research Site, Torrance, California
  - Research Site, Fort Collins, Colorado
  - Research Site, Danbury, Connecticut
  - Research Site, Hartford, Connecticut
  - Research Site, Newark, Delaware
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Atlantis, Florida
  - Research Site, Daytona Beach, Florida
  - Research Site, Fort Lauderdale, Florida
  - Research Site, Hollywood, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Jupiter, Florida
  - Research Site, Melbourne, Florida
  - Research Site, Miami Beach, Florida
  - Research Site, Ocala, Florida
  - Research Site, Orlando, Florida
  - Research Site, Ormond Beach, Florida
  - Research Site, Pensacola, Florida
  - Research Site, Sarasota, Florida
  - Research Site, St. Petersburg, Florida
  - Research Site, Chicago, Illinois
  - Research Site, Park Ridge, Illinois
  - Research Site, Rock Island, Illinois
  - Research Site, Rockford, Illinois
  - Research Site, Indianapolis, Indiana
  - Research Site, Muncie, Indiana
  - Research Site, Valparaiso, Indiana
  - Research Site, Iowa City, Iowa
  - Research Site, West Des Moines, Iowa
  - Research Site, Kansas City, Kansas
  - Research Site, Olathe, Kansas
  - Research Site, Ashland, Kentucky
  - Research Site, Louisville, Kentucky
  - Research Site, Shreveport, Louisiana
  - Research Site, Auburn, Maine
  - Research Site, Bangor, Maine
  - Research Site, Baltimore, Maryland
  - Research Site, Bethesda, Maryland
  - Research Site, Salisbury, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, Springfield, Massachusetts
  - Research Site, Ann Arbor, Michigan
  - Research Site, Kalamazoo, Michigan
  - Research Site, Lansing, Michigan
  - Research Site, Laper, Michigan
  - Research Site, Pontiac, Michigan
  - Research Site, Royal Oak, Michigan
  - Research Site, Saginaw, Michigan
  - Research Site, Troy, Michigan
  - Research Site, Ypsilanti, Michigan
  - Research Site, Duluth, Minnesota
  - Research Site, Minneapolis, Minnesota
  - Research Site, Saint Paul, Minnesota
  - Research Site, Tupelo, Mississippi
  - Research Site, Columbia, Missouri
  - Research Site, Joplin, Missouri
  - Research Site, Kansas City, Missouri
  - Research Site, St Louis, Missouri
  - Research Site, Lincoln, Nebraska
  - Research Site, Omaha, Nebraska
  - Research Site, Papillion, Nebraska
  - Research Site, Newark, New Jersey
  - Research Site, Oakland, New Jersey
  - Research Site, Paterson, New Jersey
  - Research Site, Albuquerque, New Mexico
  - Research Site, Brooklyn, New York
  - Research Site, Buffalo, New York
  - Research Site, Johnson City, New York
  - Research Site, Kingston, New York
  - Research Site, New Hartford, New York
  - Research Site, New York, New York
  - Research Site, Rochester, New York
  - Research Site, Syracuse, New York
  - Research Site, Williamsville, New York
  - Research Site, Chapel Hill, North Carolina
  - Research Site, Charlotte, North Carolina
  - Research Site, Greensboro, North Carolina
  - Research Site, High Point, North Carolina
  - Research Site, Raleigh, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Cleveland, Ohio
  - Research Site, Columbus, Ohio
  - Research Site, Kettering, Ohio
  - Research Site, Zanesville, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Tulsa, Oklahoma
  - Research Site, Bend, Oregon
  - Research Site, Camp Hill, Pennsylvania
  - Research Site, Danville, Pennsylvania
  - Research Site, Doylestown, Pennsylvania
  - Research Site, Harrisburg, Pennsylvania
  - Research Site, Lancaster, Pennsylvania
  - Research Site, Langhorne, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Sayre, Pennsylvania
  - Research Site, Sellersville, Pennsylvania
  - Research Site, Wormleysburg, Pennsylvania
  - Research Site, York, Pennsylvania
  - Research Site, Providence, Rhode Island
  - Research Site, Wakefield, Rhode Island
  - Research Site, Anderson, South Carolina
  - Research Site, Charleston, South Carolina
  - Research Site, Columbia, South Carolina
  - Research Site, Greenville, South Carolina
  - Research Site, Rapid City, South Dakota
  - Research Site, Jackson, Tennessee
  - Research Site, Knoxville, Tennessee
  - Research Site, Memphis, Tennessee
  - Research Site, Amarillo, Texas
  - Research Site, Austin, Texas
  - Research Site, Dallas, Texas
  - Research Site, Houston, Texas
  - Research Site, Lubbock, Texas
  - Research Site, San Antonio, Texas
  - Research Site, San Marcos, Texas
  - Research Site, Tyler, Texas
  - Research Site, Victoria, Texas
  - Research Site, Burlington, Vermont
  - Research Site, Falls Church, Virginia
  - Research Site, Fredericksburg, Virginia
  - Research Site, Norfolk, Virginia
  - Research Site, Winchester, Virginia
  - Research Site, Everett, Washington
  - Research Site, Tacoma, Washington
  - Research Site, Morgantown, West Virginia
  - Research Site, Green Bay, Wisconsin
- Argentina (13):
  - Research Site, Adrogué, Buenos Aires
  - Research Site, Buenos Aires, Buenos Aires
  - Research Site, Capital Federal, Buenos Aires
  - Research Site, Ciudad Autonoma de Bs. As., Buenos Aires
  - Research Site, Quilmes, Buenos Aires
  - Research Site, Corrientes, Corrientes Province
  - Research Site, Córdoba, Córdoba Province
  - Research Site, Morón, Pcia. de Buenos Aires
  - Research Site, Salta, Salta Province
  - Research Site, Rosario, Santa Fe Province
  - Research Site, Santa Fe, Santa Fe Province
  - Research Site, San Miguel de Tucumán, Tucuman - Argentina
  - Research Site, San Miguel de Tucumán
- Australia (9):
  - Research Site, Bruce, Australian Capital Territory
  - Research Site, Chermside, Queensland
  - Research Site, Herston, Queensland
  - Research Site, Woolloongabba, Queensland
  - Research Site, Bedford Park, South Australia
  - Research Site, Dandenong, Victoria
  - Research Site, Geelong, Victoria
  - Research Site, Melbourne, Victoria
  - Research Site, Perth, Western Australia
- Austria (8):
  - Research Site, Feldkirch
  - Research Site, Freistadt
  - Research Site, Graz
  - Research Site, Innsbruck
  - Research Site, Linz
  - Research Site, Mödling
  - Research Site, Vienna
  - Research Site, Villach
- Belgium (13):
  - Research Site, Aalst, Belgium
  - Research Site, Bouge, Belgium
  - Research Site, Brasschaat, Belgium
  - Research Site, Brussels (anderlecht), Belgium
  - Research Site, Charleroi, Belgium
  - Research Site, Edegem, Belgium
  - Research Site, Genk, Belgium
  - Research Site, Hasselt, Belgium
  - Research Site, Huy, Belgium
  - Research Site, Liège, Belgium
  - Research Site, Mechelen, Belgium
  - Research Site, Mol, Belgium
  - Research Site, Wilrijk, Belgium
- Brazil (18):
  - Research Site, Maceió, Alagoas
  - Research Site, Salvador, Estado de Bahia
  - Research Site, Brasília, Federal District
  - Research Site, Goiânia, Goiás
  - Research Site, Campo Grande, Mato Grosso do Sul
  - Research Site, Belo Horizonte, Minas Gerais
  - Research Site, Uberlândia, Minas Gerais
  - Research Site, Curitiba, Paraná
  - Research Site, Maringá, Paraná
  - Research Site, Recife, Pernambuco
  - Research Site, Rio de Janeiro, Rio de Janeiro
  - Research Site, Natal, Rio Grande do Norte
  - Research Site, Porto Alegre, Rio Grande do Sul
  - Research Site, São José, Santa Catarina
  - Research Site, Aracaju, Sergipe
  - Research Site, S.j.rio Preto, São Paulo
  - Research Site, São Paulo, São Paulo
  - Research Site, Campinas
- Bulgaria (11):
  - Research Site, Burgas
  - Research Site, Dimitrovgrad
  - Research Site, Gabrovo
  - Research Site, Haskovo
  - Research Site, Kazanlak
  - Research Site, Pleven
  - Research Site, Plovdiv
  - Research Site, Rousse
  - Research Site, Smolyan
  - Research Site, Sofia
  - Research Site, Varna
- Canada (28):
  - Research Site, Calgary, Alberta
  - Research Site, Edmonton, Alberta
  - Research Site, Campbell River, British Columbia
  - Research Site, Kelowna, British Columbia
  - Research Site, New Westminster, British Columbia
  - Research Site, Penticton, British Columbia
  - Research Site, Surrey, British Columbia
  - Research Site, Vancouver, British Columbia
  - Research Site, Victoria, British Columbia
  - Research Site, Winnipeg, Manitoba
  - Research Site, Saint John, New Brunswick
  - Research Site, St. John's, Newfoundland and Labrador
  - Research Site, Brockville, Ontario
  - Research Site, Cambridge, Ontario
  - Research Site, Cornwall, Ontario
  - Research Site, London, Ontario
  - Research Site, Newmarket, Ontario
  - Research Site, Oshawa, Ontario
  - Research Site, Ottawa, Ontario
  - Research Site, Scarborough Village, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Laval, Quebec
  - Research Site, Montreal, Quebec
  - Research Site, Québec, Quebec
  - Research Site, Saint-Georges, Quebec
  - Research Site, Sherbrooke, Quebec
  - Research Site, Thetford-Mines, Quebec
  - Research Site, Regina, Saskatchewan
- China (6):
  - Research Site, Beijing, China
  - Research Site, Shanghai, Pudong, China
  - Research Site, Guangzhou, Guangdong
  - Research Site, Shenyang, Liaoning
  - Research Site, Chengdu, Sichuan
  - Research Site, Hangzhou
- Czechia (15):
  - Research Site, Brno, CZ
  - Research Site, Hradec Králové
  - Research Site, Jihlava
  - Research Site, Kladno
  - Research Site, Liberec
  - Research Site, Olomouc
  - Research Site, Ostrava-poruba
  - Research Site, Pardubice
  - Research Site, Prague
  - Research Site, Slaný
  - Research Site, Teplice
  - Research Site, Ústí nad Labem
  - Research Site, Ústí nad Orlicí
  - Research Site, Zlín
  - Research Site, Znojmo
- Denmark (22):
  - Research Site, Copenhagen
  - Research Site, Esbjerg
  - Research Site, Fredericia
  - Research Site, Frederiksberg
  - Research Site, Frederikssund
  - Research Site, Glostrup Municipality
  - Research Site, Hellerup
  - Research Site, Herlev
  - Research Site, Herning
  - Research Site, Hillerød
  - Research Site, Hjørring
  - Research Site, Holbæk
  - Research Site, Horsens
  - Research Site, Hvidovre
  - Research Site, Kolding
  - Research Site, Køge
  - Research Site, Næstved
  - Research Site, Odense C
  - Research Site, Roskilde
  - Research Site, Silkeborg
  - Research Site, Slagelse
  - Research Site, Viborg
- Finland (9):
  - Research Site, Kokkola, Finland
  - Research Site, Rovaniemi, Finland
  - Research Site, Turku, Finland
  - Research Site, Hus (helsinki)
  - Research Site, Jyväskylä
  - Research Site, Kuopio
  - Research Site, Lahti
  - Research Site, Lappeenranta
  - Research Site, Pori
- France (34):
  - Research Site, Abbeville
  - Research Site, Allauch
  - Research Site, Arras
  - Research Site, Avignon
  - Research Site, Bayonne
  - Research Site, Besançon
  - Research Site, Brest
  - Research Site, Caen
  - Research Site, Cholet
  - Research Site, Créteil
  - Research Site, Croix
  - Research Site, Dijon
  - Research Site, Douai
  - Research Site, Falaise
  - Research Site, Fréjus
  - Research Site, La Rochelle
  - Research Site, Lagny-sur-Marne
  - Research Site, Lille
  - Research Site, Limoges
  - Research Site, Lomme
  - Research Site, Marseille
  - Research Site, Nîmes
  - Research Site, Orléans
  - Research Site, Paris
  - Research Site, Pau
  - Research Site, Pessac
  - Research Site, Quincy-sous-Sénart
  - Research Site, Rennes
  - Research Site, Rouen
  - Research Site, Senlis
  - Research Site, Strasbourg
  - Research Site, Toulouse
  - Research Site, Tourcoing
  - Research Site, Valenciennes
- Research Site, Tbilisi, Georgia
- Germany (39):
  - Research Site, Aschaffenburg
  - Research Site, Bad Mergentheim
  - Research Site, Bad Nauheim
  - Research Site, Bad Rothenfelde
  - Research Site, Berlin
  - Research Site, Bochum
  - Research Site, Bonn
  - Research Site, Cloppenburg
  - Research Site, Coburg
  - Research Site, Dortmund
  - Research Site, Dresden
  - Research Site, Duisburg
  - Research Site, Erfurt
  - Research Site, Essen
  - Research Site, Esslingen am Neckar
  - Research Site, Frankfurt
  - Research Site, Göttingen
  - Research Site, Greifswald
  - Research Site, Halle
  - Research Site, Hamburg
  - Research Site, Hanover
  - Research Site, Heidelberg
  - Research Site, Jena
  - Research Site, Kiel
  - Research Site, Krefeld
  - Research Site, Limburg
  - Research Site, Lübeck
  - Research Site, Mainz
  - Research Site, Merseburg
  - Research Site, Mönchengladbach
  - Research Site, Muhlheim An Der Ruhr
  - Research Site, Münster
  - Research Site, Regensburg
  - Research Site, Rostock
  - Research Site, Ulm
  - Research Site, Warendorf
  - Research Site, Witten
  - Research Site, Wuppertal
  - Research Site, Würzburg
- Greece (6):
  - Research Site, Heraklion, Crete
  - Research Site, Athens, Greece
  - Research Site, Larissa, Greece
  - Research Site, Piraeus, Greece
  - Research Site, Thessaloniki, Greece
  - Research Site, Pátrai
- Research Site, Hong Kong, Hong Kong
- Hungary (11):
  - Research Site, Budapest
  - Research Site, Cegléd
  - Research Site, Debrecen
  - Research Site, Gyula
  - Research Site, Hodmez-vasarhely
  - Research Site, Kaposvár
  - Research Site, Kecskemét
  - Research Site, Mosonmagyaróvár
  - Research Site, Pécs
  - Research Site, Székesfehérvár
  - Research Site, Zalaegerszeg
- India (18):
  - Research Site, Hyderabad, Andhrapradesh
  - Research Site, Vijayawada, Andhrapradesh
  - Research Site, Ahmedabad, Gujarat
  - Research Site, Gandhinagar, Gujarat
  - Research Site, Vadodara, Gujarat
  - Research Site, Bangalore, Karnataka
  - Research Site, Kochi, Kerala
  - Research Site, Thrissur, Kerala
  - Research Site, Bhopal, Madhya Pradesh
  - Research Site, Mumbai, Maharashtra
  - Research Site, Nagpur, Maharashtra
  - Research Site, New Delhi, National Capital Territory of Delhi
  - Research Site, Patiāla, Punjab
  - Research Site, Bikaner, Rajasthan
  - Research Site, Jaipur, Rajasthan
  - Research Site, Chennai, Tamil Nadu
  - Research Site, Coimabatore, Tamil Nadu
  - Research Site, Kolkata, West Bengal
- Indonesia (6):
  - Research Site, Denpasar, Bali
  - Research Site, Surabaya, East Java
  - Research Site, Bandung, West Java
  - Research Site, Jakarta
  - Research Site, Makassar
  - Research Site, Semarang
- Israel (11):
  - Research Site, Afula
  - Research Site, Ashkelon
  - Research Site, Beersheba
  - Research Site, Hadera
  - Research Site, Haifa
  - Research Site, Holon
  - Research Site, Jerusalem
  - Research Site, Poriya M.p. Lower Galilee
  - Research Site, Rehovot
  - Research Site, Tel Aviv
  - Research Site, Ẕerifin
- Italy (29):
  - Research Site, Ancona, AN
  - Research Site, Bari, BA
  - Research Site, Bergamo, BG
  - Research Site, Caserta, CE
  - Research Site, Catania, CT
  - Research Site, Ferrara, FE
  - Research Site, Foggia, FG
  - Research Site, San Giovanni Rotondo, FG
  - Research Site, Bagno a Ripoli, FI
  - Research Site, Florence, FI
  - Research Site, Legnano, MI
  - Research Site, Milan, MI
  - Research Site, Monza, MI
  - Research Site, Rozzano, MI
  - Research Site, Mantova, MN
  - Research Site, Modena, MO
  - Research Site, Pescara, PE
  - Research Site, Parma, PR
  - Research Site, Pavia, PV
  - Research Site, Lido di Ostia, Roma
  - Research Site, Sassari, SS
  - Research Site, Treviso, TV
  - Research Site, Varese, VA
  - Research Site, Mestre, VE
  - Research Site, Verona, VR
  - Research Site, Massa Carrara
  - Research Site, Napoli
  - Research Site, Novara
  - Research Site, Roma
- Malaysia (3):
  - Research Site, Kuala Lumpur, Kuala Lumpur
  - Research Site, Kuching, Sarawak
  - Research Site, George Town
- Mexico (6):
  - Research Site, Durango, Durango
  - Research Site, Guadalajara, Jalisco
  - Research Site, Zapopan, Jalisco
  - Research Site, Mexico City, Mexico City
  - Research Site, Monterrey, Nuevo León
  - Research Site, Puebla City, Puebla
- Netherlands (36):
  - Research Site, Alkmaar
  - Research Site, Almelo
  - Research Site, Amersfoort
  - Research Site, Amsterdam
  - Research Site, Apeldoorn
  - Research Site, Arnhem
  - Research Site, Assen
  - Research Site, Blaricum
  - Research Site, Breda
  - Research Site, Capelle aan den IJssel
  - Research Site, Delft
  - Research Site, Deventer
  - Research Site, Dordrecht
  - Research Site, Drachten
  - Research Site, Ede
  - Research Site, Eindhoven
  - Research Site, Goes
  - Research Site, Gorinchem
  - Research Site, Gouda
  - Research Site, Haarlem
  - Research Site, Hardenberg
  - Research Site, Harderwijk
  - Research Site, Heerlen
  - Research Site, Helmond
  - Research Site, Hilversum
  - Research Site, Leeuwarden
  - Research Site, Maastricht
  - Research Site, Nieuwegein
  - Research Site, Nijmegen
  - Research Site, Rotterdam
  - Research Site, Spijkenisse
  - Research Site, The Hague
  - Research Site, Tiel
  - Research Site, Tilburg
  - Research Site, Veldhoven
  - Research Site, Vlaardingen
- Norway (16):
  - Research Site, Arendal
  - Research Site, Bergen
  - Research Site, Bodø
  - Research Site, Drammen
  - Research Site, Flekkefjord
  - Research Site, Gjøvik
  - Research Site, Hamar
  - Research Site, Kongsberg
  - Research Site, Kristiansand
  - Research Site, Lillehammer
  - Research Site, Nordbyhagen
  - Research Site, Notodden
  - Research Site, Oslo
  - Research Site, Rud
  - Research Site, Tromsø
  - Research Site, Tynset
- Philippines (5):
  - Research Site, Pasig, Philippines
  - Research Site, Cebu
  - Research Site, Davao City
  - Research Site, Manila
  - Research Site, Quezon City
- Poland (30):
  - Research Site, Bialystok
  - Research Site, Bielsko-Biala
  - Research Site, Bydgoszcz
  - Research Site, Bytom
  - Research Site, Częstochowa
  - Research Site, Elblag
  - Research Site, Gda?sk
  - Research Site, Gdynia
  - Research Site, Grodzisk Mazowiecki
  - Research Site, Inowrocław
  - Research Site, Katowice
  - Research Site, Krakow
  - Research Site, Lodz
  - Research Site, Lublin
  - Research Site, Olsztyn
  - Research Site, Opole
  - Research Site, Ostrowiec Świętokrzyski
  - Research Site, Oława
  - Research Site, Poznan
  - Research Site, Płock
  - Research Site, Radom
  - Research Site, Szczecin
  - Research Site, Tarnów
  - Research Site, Torun
  - Research Site, Warsaw
  - Research Site, Wałbrzych
  - Research Site, Wejherowo
  - Research Site, Wroclaw
  - Research Site, Włocławek
  - Research Site, Zamość
- Portugal (12):
  - Research Site, Amadora
  - Research Site, Aveiro
  - Research Site, Braga
  - Research Site, Coimbra
  - Research Site, Leiria
  - Research Site, Lisbon
  - Research Site, Penafiel
  - Research Site, Santa Maria da Feira
  - Research Site, Santarém
  - Research Site, Setúbal
  - Research Site, Vila Nova de Gaia
  - Research Site, Vila Real
- Research Site, San Juan, Puerto Rico
- Romania (10):
  - Research Site, Piteşti, Argeş
  - Research Site, Brasov, Brașov County
  - Research Site, Brăila, Brăila County
  - Research Site, Cluj-Napoca, Cluj
  - Research Site, Iași, Iaşi
  - Research Site, Bucharest
  - Research Site, Buzău
  - Research Site, Craiova
  - Research Site, Iași
  - Research Site, Suceava
- Russia (19):
  - Research Site, Khanty-Mansiysk, Khanty-mansiysk Autonomous Dis
  - Research Site, Barnaul
  - Research Site, Irkutsk
  - Research Site, Kaliningrad
  - Research Site, Kazan'
  - Research Site, Kemerovo
  - Research Site, Krasnodar
  - Research Site, Krasnoyarsk
  - Research Site, Moscow
  - Research Site, Murmansk
  - Research Site, Nizhny Novgorod
  - Research Site, Novosibirsk
  - Research Site, Rostov-on-Don
  - Research Site, Saint Petersburg
  - Research Site, Samara
  - Research Site, Tomsk
  - Research Site, Tyumen
  - Research Site, Vladivostok
  - Research Site, Yekaterinburg
- Research Site, Singapore, Singapore, Singapore
- Slovakia (10):
  - Research Site, Bratislava
  - Research Site, Košice
  - Research Site, Liptovský Mikuláš
  - Research Site, Martin
  - Research Site, Nitra
  - Research Site, Nové Zámky
  - Research Site, Piešťany
  - Research Site, Ružomberok
  - Research Site, Trnava
  - Research Site, Žilina
- South Africa (4):
  - Research Site, Cape Town, Cape Town
  - Research Site, Somerset West, Cape Town
  - Research Site, Bloemfontein, Free State
  - Research Site, Pretoria
- South Korea (6):
  - Research Site, Seongnam, Gyeonggido
  - Research Site, Daegu
  - Research Site, Gwangju
  - Research Site, Seoul
  - Research Site, Suwon
  - Research Site, Wŏnju
- Spain (11):
  - Research Site, Málaga, Andalusia
  - Research Site, Seville, Andalusia
  - Research Site, Palma de Mallorca, Balearic Islands
  - Research Site, Barcelona, Catalonia
  - Research Site, Lleida, Catalonia
  - Research Site, Terrassa, Catalonia
  - Research Site, Cáceres, Extremadura
  - Research Site, Vigo(pontevedra), Galicia
  - Research Site, Madrid, Madrid
  - Research Site, Gijón, Principality of Asturias
  - Research Site, Valencia, Valencia
- Sweden (18):
  - Research Site, Borås
  - Research Site, Eksjö
  - Research Site, Eskilstuna
  - Research Site, Falun
  - Research Site, Halmstad
  - Research Site, Jönköping
  - Research Site, Kalmar
  - Research Site, Karlskrona
  - Research Site, Lidköping
  - Research Site, Linköping
  - Research Site, Ljungby
  - Research Site, Lund
  - Research Site, Östersund
  - Research Site, Skövde
  - Research Site, Stockholm
  - Research Site, Sundsvall
  - Research Site, Uppsala
  - Research Site, Västerås
- Switzerland (6):
  - Research Site, Mendrisio, Canton Ticino
  - Research Site, Bellinzona
  - Research Site, Bern
  - Research Site, Geneva
  - Research Site, Kreuzlingen
  - Research Site, Lugano
- Taiwan (3):
  - Research Site, Niao-song-shiang, Kaohsiung
  - Research Site, Kweishan Shiang, Taoyuan Hsien
  - Research Site, Taipei
- Thailand (3):
  - Research Site, Bangkok, Bangkok
  - Research Site, Chiang Mai, Thailand
  - Research Site, Khon Kaen, Thailand
- Turkey (Türkiye) (5):
  - Research Site, Istanbul, Kartal
  - Research Site, Ankara, Sihhiye
  - Research Site, Adana
  - Research Site, Antalya
  - Research Site, Mersin
- Ukraine (5):
  - Research Site, Dnipro
  - Research Site, Donetsk
  - Research Site, Kharkiv
  - Research Site, Kiev
  - Research Site, Makiyivka
- United Kingdom (15):
  - Research Site, Airdrie, Lanarkshire
  - Research Site, Belfast, Northern Ireland
  - Research Site, Basingstoke
  - Research Site, Birmingham
  - Research Site, Blackpool
  - Research Site, Dundee
  - Research Site, Edinburgh
  - Research Site, Glasgow
  - Research Site, Leicester
  - Research Site, London
  - Research Site, Manchester
  - Research Site, Middlesbrough
  - Research Site, Poole
  - Research Site, Sheffield
  - Research Site, Swansea

REFERENCES:
- [Derived] Serebruany VL, Tanguay JF, Gurvich ML, Marciniak TA, Atar D. Strokes and Transient Ischemic Attacks Occurrence During Annual Dual Antiplatelet Therapy. Am J Ther. 2023 Sep-Oct 01;30(5):e411-e415. doi: 10.1097/MJT.0000000000001622. Epub 2023 Mar 29. PMID 37713684
- [Derived] Hjort M, Eggers KM, Lakic TG, Lindback J, Budaj A, Cornel JH, Giannitsis E, Katus HA, Siegbahn A, Storey RF, Becker RC, Wallentin L, Lindahl B; PLATO trial investigators*. Biomarker Concentrations and Their Temporal Changes in Patients With Myocardial Infarction and Nonobstructive Compared With Obstructive Coronary Arteries: Results From the PLATO Trial. J Am Heart Assoc. 2023 Jan 3;12(1):e027466. doi: 10.1161/JAHA.122.027466. Epub 2022 Dec 24. PMID 36565198
- [Derived] Batra G, Lindback J, Becker RC, Harrington RA, Held C, James SK, Kempf T, Lopes RD, Mahaffey KW, Steg PG, Storey RF, Swahn E, Wollert KC, Siegbahn A, Wallentin L. Biomarker-Based Prediction of Recurrent Ischemic Events in Patients With Acute Coronary Syndromes. J Am Coll Cardiol. 2022 Nov 1;80(18):1735-1747. doi: 10.1016/j.jacc.2022.08.767. PMID 36302586
- [Derived] Natale P, Palmer SC, Saglimbene VM, Ruospo M, Razavian M, Craig JC, Jardine MJ, Webster AC, Strippoli GF. Antiplatelet agents for chronic kidney disease. Cochrane Database Syst Rev. 2022 Feb 28;2(2):CD008834. doi: 10.1002/14651858.CD008834.pub4. PMID 35224730
- [Derived] Samman KN, Mehanna P, Takla E, Grenier JC, Chan MY, Lopes RD, Neely ML, Wang TY, Newby LK, Becker RC, Lordkipanidze M, Ruiz M, Hussin JG, Jolicoeur EM. Differential modulation of polyunsaturated fatty acids in patients with myocardial infarction treated with ticagrelor or clopidogrel. Cell Rep Med. 2021 Jun 4;2(6):100299. doi: 10.1016/j.xcrm.2021.100299. eCollection 2021 Jun 15. PMID 34195679
- [Derived] Thi Thu Nguyen T, Van Do D, Mellstrom C, Quang Nguyen T, Manh Pham H, Van Hoang S, Cong Luu T, Le Phuong T. Cost-Effectiveness of Ticagrelor Compared with Clopidogrel in Patients with Acute Coronary Syndrome from Vietnamese Healthcare Payers' Perspective. Adv Ther. 2021 Jul;38(7):4026-4039. doi: 10.1007/s12325-021-01743-5. Epub 2021 Jun 11. PMID 34115329
- [Derived] Mahmoodi BK, Eriksson N, Vos GJA, Meijer K, Siegbahn A, James S, Wallentin L, Ten Berg JM. Factor V Leiden Does Not Modify the Phenotype of Acute Coronary Syndrome or the Extent of Myocardial Necrosis. J Am Heart Assoc. 2021 Jun;10(11):e020025. doi: 10.1161/JAHA.120.020025. Epub 2021 May 17. PMID 33998271
- [Derived] Gregersen I, Michelsen AE, Lunde NN, Akerblom A, Lakic TG, Skjelland M, Ryeng Skagen K, Becker RC, Lindback J, Himmelmann A, Solberg R, Johansen HT, James SK, Siegbahn A, Storey RF, Kontny F, Aukrust P, Ueland T, Wallentin L, Halvorsen B. Legumain in Acute Coronary Syndromes: A Substudy of the PLATO (Platelet Inhibition and Patient Outcomes) Trial. J Am Heart Assoc. 2020 Sep;9(17):e016360. doi: 10.1161/JAHA.120.016360. Epub 2020 Aug 15. PMID 32809893
- [Derived] Sumaya W, Wallentin L, James SK, Siegbahn A, Gabrysch K, Himmelmann A, Ajjan RA, Storey RF. Impaired Fibrinolysis Predicts Adverse Outcome in Acute Coronary Syndrome Patients with Diabetes: A PLATO Sub-Study. Thromb Haemost. 2020 Mar;120(3):412-422. doi: 10.1055/s-0039-1701011. Epub 2020 Jan 23. PMID 31975352
- [Derived] Ueland T, Akerblom A, Ghukasyan T, Michelsen AE, Becker RC, Bertilsson M, Budaj A, Cornel JH, Himmelmann A, James SK, Siegbahn A, Storey RF, Kontny F, Aukrust P, Wallentin L; PLATO Investigators. ALCAM predicts future cardiovascular death in acute coronary syndromes: Insights from the PLATO trial. Atherosclerosis. 2020 Jan;293:35-41. doi: 10.1016/j.atherosclerosis.2019.11.031. Epub 2019 Nov 29. PMID 31835039
- [Derived] Andersen T, Ueland T, Ghukasyan Lakic T, Akerblom A, Bertilsson M, Aukrust P, Michelsen AE, James SK, Becker RC, Storey RF, Wallentin L, Siegbahn A, Kontny F. C-X-C Ligand 16 Is an Independent Predictor of Cardiovascular Death and Morbidity in Acute Coronary Syndromes. Arterioscler Thromb Vasc Biol. 2019 Nov;39(11):2402-2410. doi: 10.1161/ATVBAHA.119.312633. Epub 2019 Sep 26. PMID 31554419
- [Derived] Akerblom A, Wojdyla DM, Wallentin L, James SK, de Souza Brito F, Steg PG, Cannon CP, Katus HA, Himmelmann A, Storey RF, Becker RC, Lopes RD; PLATO Investigators. Ticagrelor in patients with heart failure after acute coronary syndromes-Insights from the PLATelet inhibition and patient Outcomes (PLATO) trial. Am Heart J. 2019 Jul;213:57-65. doi: 10.1016/j.ahj.2019.04.006. Epub 2019 Apr 18. PMID 31108273
- [Derived] Franchi F, James SK, Ghukasyan Lakic T, Budaj AJ, Cornel JH, Katus HA, Keltai M, Kontny F, Lewis BS, Storey RF, Himmelmann A, Wallentin L, Angiolillo DJ; PLATO Investigators. Impact of Diabetes Mellitus and Chronic Kidney Disease on Cardiovascular Outcomes and Platelet P2Y12 Receptor Antagonist Effects in Patients With Acute Coronary Syndromes: Insights From the PLATO Trial. J Am Heart Assoc. 2019 Mar 19;8(6):e011139. doi: 10.1161/JAHA.118.011139. PMID 30857464
- [Derived] Lindholm D, James SK, Gabrysch K, Storey RF, Himmelmann A, Cannon CP, Mahaffey KW, Steg PG, Held C, Siegbahn A, Wallentin L. Association of Multiple Biomarkers With Risk of All-Cause and Cause-Specific Mortality After Acute Coronary Syndromes: A Secondary Analysis of the PLATO Biomarker Study. JAMA Cardiol. 2018 Dec 1;3(12):1160-1166. doi: 10.1001/jamacardio.2018.3811. PMID 30427997
- [Derived] Inohara T, Pieper K, Wojdyla DM, Patel MR, Jones WS, Tricoci P, Mahaffey KW, James SK, Alexander JH, Lopes RD, Wallentin L, Ohman EM, Roe MT, Vemulapalli S. Incidence, timing, and type of first and recurrent ischemic events in patients with and without peripheral artery disease after an acute coronary syndrome. Am Heart J. 2018 Jul;201:25-32. doi: 10.1016/j.ahj.2018.03.013. Epub 2018 Mar 28. PMID 29910052
- [Derived] Ueland T, Akerblom A, Ghukasyan T, Michelsen AE, Aukrust P, Becker RC, Bertilsson M, Himmelmann A, James SK, Siegbahn A, Storey RF, Kontny F, Wallentin L; PLATO (Platelet Inhibition and Patient Outcomes) Trial Investigators. Osteoprotegerin Is Associated With Major Bleeding But Not With Cardiovascular Outcomes in Patients With Acute Coronary Syndromes: Insights From the PLATO (Platelet Inhibition and Patient Outcomes) Trial. J Am Heart Assoc. 2018 Jan 12;7(2):e007009. doi: 10.1161/JAHA.117.007009. PMID 29330256
- [Derived] Bellavia A, Wallentin L, Orsini N, James SK, Cannon CP, Himmelmann A, Sundstrom J, Renlund H, Lytsy P. Time-based measures of treatment effect: reassessment of ticagrelor and clopidogrel from the PLATO trial. Open Heart. 2017 Jun 1;4(2):e000557. doi: 10.1136/openhrt-2016-000557. eCollection 2017. PMID 28761675
- [Derived] Lindholm D, Hagstrom E, James SK, Becker RC, Cannon CP, Himmelmann A, Katus HA, Maurer G, Lopez-Sendon JL, Steg PG, Storey RF, Siegbahn A, Wallentin L. Growth Differentiation Factor 15 at 1 Month After an Acute Coronary Syndrome Is Associated With Increased Risk of Major Bleeding. J Am Heart Assoc. 2017 Apr 14;6(4):e005580. doi: 10.1161/JAHA.117.005580. PMID 28411246
- [Derived] Lindholm D, James SK, Bertilsson M, Becker RC, Cannon CP, Giannitsis E, Harrington RA, Himmelmann A, Kontny F, Siegbahn A, Steg PG, Storey RF, Velders MA, Weaver WD, Wallentin L; PLATO Investigators. Biomarkers and Coronary Lesions Predict Outcomes after Revascularization in Non-ST-Elevation Acute Coronary Syndrome. Clin Chem. 2017 Feb;63(2):573-584. doi: 10.1373/clinchem.2016.261271. Epub 2016 Dec 8. PMID 27932413
- [Derived] Held P, Himmelmann A, Ditmarsch M. Ticagrelor for the treatment of atherosclerotic disease: insights from the PARTHENON clinical development program. Future Cardiol. 2016 Jul;12(4):405-18. doi: 10.2217/fca-2016-0028. Epub 2016 May 10. PMID 27160944
- [Derived] Johansson A, Eriksson N, Lindholm D, Varenhorst C, James S, Syvanen AC, Axelsson T, Siegbahn A, Barratt BJ, Becker RC, Himmelmann A, Katus HA, Steg PG, Storey RF, Wallentin L; PLATO Investigators. Genome-wide association and Mendelian randomization study of NT-proBNP in patients with acute coronary syndrome. Hum Mol Genet. 2016 Apr 1;25(7):1447-56. doi: 10.1093/hmg/ddw012. Epub 2016 Jan 21. PMID 26908625
- [Derived] Velders MA, Abtan J, Angiolillo DJ, Ardissino D, Harrington RA, Hellkamp A, Himmelmann A, Husted S, Katus HA, Meier B, Schulte PJ, Storey RF, Wallentin L, Gabriel Steg P, James SK; PLATO Investigators. Safety and efficacy of ticagrelor and clopidogrel in primary percutaneous coronary intervention. Heart. 2016 Apr;102(8):617-25. doi: 10.1136/heartjnl-2015-308963. Epub 2016 Feb 4. PMID 26848185
- [Derived] Bui AH, Cannon CP, Steg PG, Storey RF, Husted S, Guo J, Im K, James SK, Michelson EL, Himmelmann A, Held C, Varenhorst C, Wallentin L, Scirica BM. Relationship Between Early and Late Nonsustained Ventricular Tachycardia and Cardiovascular Death in Patients With Acute Coronary Syndrome in the Platelet Inhibition and Patient Outcomes (PLATO) Trial. Circ Arrhythm Electrophysiol. 2016 Feb;9(2):e002951. doi: 10.1161/CIRCEP.115.002951. PMID 26810596
- [Derived] Andell P, James SK, Cannon CP, Cyr DD, Himmelmann A, Husted S, Keltai M, Koul S, Santoso A, Steg PG, Storey RF, Wallentin L, Erlinge D; PLATO Investigators. Ticagrelor Versus Clopidogrel in Patients With Acute Coronary Syndromes and Chronic Obstructive Pulmonary Disease: An Analysis From the Platelet Inhibition and Patient Outcomes (PLATO) Trial. J Am Heart Assoc. 2015 Oct 9;4(10):e002490. doi: 10.1161/JAHA.115.002490. PMID 26452988
- [Derived] Hagstrom E, James SK, Bertilsson M, Becker RC, Himmelmann A, Husted S, Katus HA, Steg PG, Storey RF, Siegbahn A, Wallentin L; PLATO Investigators. Growth differentiation factor-15 level predicts major bleeding and cardiovascular events in patients with acute coronary syndromes: results from the PLATO study. Eur Heart J. 2016 Apr 21;37(16):1325-33. doi: 10.1093/eurheartj/ehv491. Epub 2015 Sep 28. PMID 26417057
- [Derived] Mahaffey KW, Hager R, Wojdyla D, White HD, Armstrong PW, Alexander JH, Tricoci P, Lopes RD, Ohman EM, Roe MT, Harrington RA, Wallentin L. Meta-analysis of intracranial hemorrhage in acute coronary syndromes: incidence, predictors, and clinical outcomes. J Am Heart Assoc. 2015 Jun 18;4(6):e001512. doi: 10.1161/JAHA.114.001512. PMID 26089177
- [Derived] Kang HJ, Clare RM, Gao R, Held C, Himmelmann A, James SK, Lim ST, Santoso A, Yu CM, Wallentin L, Becker RC; PLATO Investigators. Ticagrelor versus clopidogrel in Asian patients with acute coronary syndrome: A retrospective analysis from the Platelet Inhibition and Patient Outcomes (PLATO) Trial. Am Heart J. 2015 Jun;169(6):899-905.e1. doi: 10.1016/j.ahj.2015.03.015. Epub 2015 Mar 31. PMID 26027629
- [Derived] Velders MA, Wallentin L, Becker RC, van Boven AJ, Himmelmann A, Husted S, Katus HA, Lindholm D, Morais J, Siegbahn A, Storey RF, Wernroth L, James SK; PLATO Investigators. Biomarkers for risk stratification of patients with ST-elevation myocardial infarction treated with primary percutaneous coronary intervention: Insights from the Platelet Inhibition and Patient Outcomes trial. Am Heart J. 2015 Jun;169(6):879-889.e7. doi: 10.1016/j.ahj.2015.02.019. Epub 2015 Mar 5. PMID 26027627
- [Derived] Varenhorst C, Eriksson N, Johansson A, Barratt BJ, Hagstrom E, Akerblom A, Syvanen AC, Becker RC, James SK, Katus HA, Husted S, Steg PG, Siegbahn A, Voora D, Teng R, Storey RF, Wallentin L; PLATO Investigators. Effect of genetic variations on ticagrelor plasma levels and clinical outcomes. Eur Heart J. 2015 Aug 1;36(29):1901-12. doi: 10.1093/eurheartj/ehv116. Epub 2015 May 2. PMID 25935875
- [Derived] Kholaif N, Zheng Y, Jagasia P, Himmelmann A, James SK, Steg PG, Storey RF, Westerhout CM, Armstrong PW. Baseline Q waves and time from symptom onset to ST-segment elevation myocardial infarction: insights from PLATO on the influence of sex. Am J Med. 2015 Aug;128(8):914.e11-9. doi: 10.1016/j.amjmed.2015.03.005. Epub 2015 Mar 26. PMID 25818495
- [Derived] Cowper PA, Pan W, Anstrom KJ, Kaul P, Wallentin L, Davidson-Ray L, Nikolic E, Janzon M, Levin LA, Cannon CP, Harrington RA, Mark DB. Economic analysis of ticagrelor therapy from a U.S. perspective: results from the PLATO study. J Am Coll Cardiol. 2015 Feb 10;65(5):465-76. doi: 10.1016/j.jacc.2014.11.034. PMID 25660925
- [Derived] Janzon M, James S, Cannon CP, Storey RF, Mellstrom C, Nicolau JC, Wallentin L, Henriksson M. Health economic analysis of ticagrelor in patients with acute coronary syndromes intended for non-invasive therapy. Heart. 2015 Jan;101(2):119-25. doi: 10.1136/heartjnl-2014-305864. Epub 2014 Sep 16. PMID 25227704
- [Derived] Varenhorst C, Alstrom U, Braun OO, Storey RF, Mahaffey KW, Bertilsson M, Cannon CP, Scirica BM, Himmelmann A, James SK, Wallentin L, Held C. Causes of mortality with ticagrelor compared with clopidogrel in acute coronary syndromes. Heart. 2014 Nov;100(22):1762-9. doi: 10.1136/heartjnl-2014-305619. Epub 2014 Jun 23. PMID 24957530
- [Derived] Kotsia A, Brilakis ES, Held C, Cannon C, Steg GP, Meier B, Cools F, Claeys MJ, Cornel JH, Aylward P, Lewis BS, Weaver D, Brandrup-Wognsen G, Stevens SR, Himmelmann A, Wallentin L, James SK. Extent of coronary artery disease and outcomes after ticagrelor administration in patients with an acute coronary syndrome: Insights from the PLATelet inhibition and patient Outcomes (PLATO) trial. Am Heart J. 2014 Jul;168(1):68-75.e2. doi: 10.1016/j.ahj.2014.04.001. Epub 2014 Apr 13. PMID 24952862
- [Derived] Patel MR, Becker RC, Wojdyla DM, Emanuelsson H, Hiatt WR, Horrow J, Husted S, Mahaffey KW, Steg PG, Storey RF, Wallentin L, James SK. Cardiovascular events in acute coronary syndrome patients with peripheral arterial disease treated with ticagrelor compared with clopidogrel: Data from the PLATO Trial. Eur J Prev Cardiol. 2015 Jun;22(6):734-42. doi: 10.1177/2047487314533215. Epub 2014 May 15. PMID 24830710
- [Derived] Husted S, James SK, Bach RG, Becker RC, Budaj A, Heras M, Himmelmann A, Horrow J, Katus HA, Lassila R, Morais J, Nicolau JC, Steg PG, Storey RF, Wojdyla D, Wallentin L; PLATO study group. The efficacy of ticagrelor is maintained in women with acute coronary syndromes participating in the prospective, randomized, PLATelet inhibition and patient Outcomes (PLATO) trial. Eur Heart J. 2014 Jun 14;35(23):1541-50. doi: 10.1093/eurheartj/ehu075. Epub 2014 Mar 28. PMID 24682844
- [Derived] Mahaffey KW, Held C, Wojdyla DM, James SK, Katus HA, Husted S, Steg PG, Cannon CP, Becker RC, Storey RF, Khurmi NS, Nicolau JC, Yu CM, Ardissino D, Budaj A, Morais J, Montgomery D, Himmelmann A, Harrington RA, Wallentin L; PLATO Investigators. Ticagrelor effects on myocardial infarction and the impact of event adjudication in the PLATO (Platelet Inhibition and Patient Outcomes) trial. J Am Coll Cardiol. 2014 Apr 22;63(15):1493-9. doi: 10.1016/j.jacc.2014.01.038. Epub 2014 Feb 19. PMID 24561148
- [Derived] Wallentin L, Lindholm D, Siegbahn A, Wernroth L, Becker RC, Cannon CP, Cornel JH, Himmelmann A, Giannitsis E, Harrington RA, Held C, Husted S, Katus HA, Mahaffey KW, Steg PG, Storey RF, James SK; PLATO study group. Biomarkers in relation to the effects of ticagrelor in comparison with clopidogrel in non-ST-elevation acute coronary syndrome patients managed with or without in-hospital revascularization: a substudy from the Prospective Randomized Platelet Inhibition and Patient Outcomes (PLATO) trial. Circulation. 2014 Jan 21;129(3):293-303. doi: 10.1161/CIRCULATIONAHA.113.004420. Epub 2013 Oct 29. PMID 24170388
- [Derived] Brilakis ES, Held C, Meier B, Cools F, Claeys MJ, Cornel JH, Aylward P, Lewis BS, Weaver D, Brandrup-Wognsen G, Stevens SR, Himmelmann A, Wallentin L, James SK. Effect of ticagrelor on the outcomes of patients with prior coronary artery bypass graft surgery: insights from the PLATelet inhibition and patient outcomes (PLATO) trial. Am Heart J. 2013 Sep;166(3):474-80. doi: 10.1016/j.ahj.2013.06.019. Epub 2013 Jul 26. PMID 24016496
- [Derived] Steg PG, Harrington RA, Emanuelsson H, Katus HA, Mahaffey KW, Meier B, Storey RF, Wojdyla DM, Lewis BS, Maurer G, Wallentin L, James SK; PLATO Study Group. Stent thrombosis with ticagrelor versus clopidogrel in patients with acute coronary syndromes: an analysis from the prospective, randomized PLATO trial. Circulation. 2013 Sep 3;128(10):1055-65. doi: 10.1161/CIRCULATIONAHA.113.002589. Epub 2013 Jul 30. PMID 23900047
- [Derived] Kunadian V, James SK, Wojdyla DM, Zorkun C, Wu J, Storey RF, Steg PG, Katus H, Emanuelsson H, Horrow J, Maya J, Wallentin L, Harrington RA, Gibson CM. Angiographic outcomes in the PLATO Trial (Platelet Inhibition and Patient Outcomes). JACC Cardiovasc Interv. 2013 Jul;6(7):671-83. doi: 10.1016/j.jcin.2013.03.014. PMID 23866179
- [Derived] James SK, Storey RF, Pieper KS, Cannon CP, Becker RC, Steg PG, Wallentin L, Harrington RA; PLATO Study Group. Response to letter regarding article, "Ticagrelor in patients with acute coronary syndromes and stroke: interpretation of subgroups in clinical trials". Stroke. 2013 Aug;44(8):e95-6. doi: 10.1161/STROKEAHA.113.002069. Epub 2013 Jun 25. No abstract available. PMID 23800556
- [Derived] James SK, Pieper KS, Cannon CP, Storey RF, Becker RC, Steg PG, Wallentin L, Harrington RA; PLATO study group. Ticagrelor in patients with acute coronary syndromes and stroke: interpretation of subgroups in clinical trials. Stroke. 2013 May;44(5):1477-9. doi: 10.1161/STROKEAHA.111.000514. Epub 2013 Apr 9. No abstract available. PMID 23572474
- [Derived] Kohli P, Wallentin L, Reyes E, Horrow J, Husted S, Angiolillo DJ, Ardissino D, Maurer G, Morais J, Nicolau JC, Oto A, Storey RF, James SK, Cannon CP. Reduction in first and recurrent cardiovascular events with ticagrelor compared with clopidogrel in the PLATO Study. Circulation. 2013 Feb 12;127(6):673-80. doi: 10.1161/CIRCULATIONAHA.112.124248. Epub 2012 Dec 31. PMID 23277305
- [Derived] Akerblom A, Wallentin L, Siegbahn A, Becker RC, Budaj A, Horrow J, Husted S, Katus H, Claeys MJ, Storey RF, Asenblad N, James SK. Outcome and causes of renal deterioration evaluated by serial cystatin C measurements in acute coronary syndrome patients -- results from the PLATelet inhibition and patient Outcomes (PLATO) study. Am Heart J. 2012 Nov;164(5):728-34. doi: 10.1016/j.ahj.2012.08.017. Epub 2012 Oct 17. PMID 23137503
- [Derived] Varenhorst C, Alstrom U, Scirica BM, Hogue CW, Asenblad N, Storey RF, Steg PG, Horrow J, Mahaffey KW, Becker RC, James S, Cannon CP, Brandrup-Wognsen G, Wallentin L, Held C. Factors contributing to the lower mortality with ticagrelor compared with clopidogrel in patients undergoing coronary artery bypass surgery. J Am Coll Cardiol. 2012 Oct 23;60(17):1623-30. doi: 10.1016/j.jacc.2012.07.021. Epub 2012 Sep 26. PMID 23021325
- [Derived] Husted S, James S, Becker RC, Horrow J, Katus H, Storey RF, Cannon CP, Heras M, Lopes RD, Morais J, Mahaffey KW, Bach RG, Wojdyla D, Wallentin L; PLATO study group. Ticagrelor versus clopidogrel in elderly patients with acute coronary syndromes: a substudy from the prospective randomized PLATelet inhibition and patient Outcomes (PLATO) trial. Circ Cardiovasc Qual Outcomes. 2012 Sep 1;5(5):680-8. doi: 10.1161/CIRCOUTCOMES.111.964395. PMID 22991347
- [Derived] Cornel JH, Becker RC, Goodman SG, Husted S, Katus H, Santoso A, Steg G, Storey RF, Vintila M, Sun JL, Horrow J, Wallentin L, Harrington R, James S. Prior smoking status, clinical outcomes, and the comparison of ticagrelor with clopidogrel in acute coronary syndromes-insights from the PLATelet inhibition and patient Outcomes (PLATO) trial. Am Heart J. 2012 Sep;164(3):334-342.e1. doi: 10.1016/j.ahj.2012.06.005. Epub 2012 Jul 26. PMID 22980299
- [Derived] Nikolic E, Janzon M, Hauch O, Wallentin L, Henriksson M; PLATO Health Economic Substudy Group. Cost-effectiveness of treating acute coronary syndrome patients with ticagrelor for 12 months: results from the PLATO study. Eur Heart J. 2013 Jan;34(3):220-8. doi: 10.1093/eurheartj/ehs149. Epub 2012 Jun 19. PMID 22719022
- [Derived] James SK, Storey RF, Khurmi NS, Husted S, Keltai M, Mahaffey KW, Maya J, Morais J, Lopes RD, Nicolau JC, Pais P, Raev D, Lopez-Sendon JL, Stevens SR, Becker RC; PLATO Study Group. Ticagrelor versus clopidogrel in patients with acute coronary syndromes and a history of stroke or transient ischemic attack. Circulation. 2012 Jun 12;125(23):2914-21. doi: 10.1161/CIRCULATIONAHA.111.082727. Epub 2012 May 9. PMID 22572911
- [Derived] Siha H, Das D, Fu Y, Zheng Y, Westerhout CM, Storey RF, James S, Wallentin L, Armstrong PW. Baseline Q waves as a prognostic modulator in patients with ST-segment elevation: insights from the PLATO trial. CMAJ. 2012 Jul 10;184(10):1135-42. doi: 10.1503/cmaj.111683. Epub 2012 Apr 30. PMID 22546885
- [Derived] Goodman SG, Clare R, Pieper KS, Nicolau JC, Storey RF, Cantor WJ, Mahaffey KW, Angiolillo DJ, Husted S, Cannon CP, James SK, Kilhamn J, Steg PG, Harrington RA, Wallentin L; Platelet Inhibition and Patient Outcomes Trial Investigators. Association of proton pump inhibitor use on cardiovascular outcomes with clopidogrel and ticagrelor: insights from the platelet inhibition and patient outcomes trial. Circulation. 2012 Feb 28;125(8):978-86. doi: 10.1161/CIRCULATIONAHA.111.032912. Epub 2012 Jan 18. PMID 22261200
- [Derived] Armstrong PW, Siha H, Fu Y, Westerhout CM, Steg PG, James SK, Storey RF, Horrow J, Katus H, Clemmensen P, Harrington RA, Wallentin L. ST-elevation acute coronary syndromes in the Platelet Inhibition and Patient Outcomes (PLATO) trial: insights from the ECG substudy. Circulation. 2012 Jan 24;125(3):514-21. doi: 10.1161/CIRCULATIONAHA.111.047530. Epub 2011 Dec 16. PMID 22179530
- [Derived] Becker RC, Bassand JP, Budaj A, Wojdyla DM, James SK, Cornel JH, French J, Held C, Horrow J, Husted S, Lopez-Sendon J, Lassila R, Mahaffey KW, Storey RF, Harrington RA, Wallentin L. Bleeding complications with the P2Y12 receptor antagonists clopidogrel and ticagrelor in the PLATelet inhibition and patient Outcomes (PLATO) trial. Eur Heart J. 2011 Dec;32(23):2933-44. doi: 10.1093/eurheartj/ehr422. Epub 2011 Nov 16. PMID 22090660
- [Derived] Mahaffey KW, Wojdyla DM, Carroll K, Becker RC, Storey RF, Angiolillo DJ, Held C, Cannon CP, James S, Pieper KS, Horrow J, Harrington RA, Wallentin L; PLATO Investigators. Ticagrelor compared with clopidogrel by geographic region in the Platelet Inhibition and Patient Outcomes (PLATO) trial. Circulation. 2011 Aug 2;124(5):544-54. doi: 10.1161/CIRCULATIONAHA.111.047498. Epub 2011 Jun 27. PMID 21709065
- [Derived] James SK, Roe MT, Cannon CP, Cornel JH, Horrow J, Husted S, Katus H, Morais J, Steg PG, Storey RF, Stevens S, Wallentin L, Harrington RA; PLATO Study Group. Ticagrelor versus clopidogrel in patients with acute coronary syndromes intended for non-invasive management: substudy from prospective randomised PLATelet inhibition and patient Outcomes (PLATO) trial. BMJ. 2011 Jun 17;342:d3527. doi: 10.1136/bmj.d3527. PMID 21685437
- [Derived] Scirica BM, Cannon CP, Emanuelsson H, Michelson EL, Harrington RA, Husted S, James S, Katus H, Pais P, Raev D, Spinar J, Steg PG, Storey RF, Wallentin L; PLATO Investigators. The incidence of bradyarrhythmias and clinical bradyarrhythmic events in patients with acute coronary syndromes treated with ticagrelor or clopidogrel in the PLATO (Platelet Inhibition and Patient Outcomes) trial: results of the continuous electrocardiographic assessment substudy. J Am Coll Cardiol. 2011 May 10;57(19):1908-16. doi: 10.1016/j.jacc.2010.11.056. PMID 21545948
- [Derived] Steg PG, James S, Harrington RA, Ardissino D, Becker RC, Cannon CP, Emanuelsson H, Finkelstein A, Husted S, Katus H, Kilhamn J, Olofsson S, Storey RF, Weaver WD, Wallentin L; PLATO Study Group. Ticagrelor versus clopidogrel in patients with ST-elevation acute coronary syndromes intended for reperfusion with primary percutaneous coronary intervention: A Platelet Inhibition and Patient Outcomes (PLATO) trial subgroup analysis. Circulation. 2010 Nov 23;122(21):2131-41. doi: 10.1161/CIRCULATIONAHA.109.927582. Epub 2010 Nov 8. PMID 21060072
- [Derived] James S, Budaj A, Aylward P, Buck KK, Cannon CP, Cornel JH, Harrington RA, Horrow J, Katus H, Keltai M, Lewis BS, Parikh K, Storey RF, Szummer K, Wojdyla D, Wallentin L. Ticagrelor versus clopidogrel in acute coronary syndromes in relation to renal function: results from the Platelet Inhibition and Patient Outcomes (PLATO) trial. Circulation. 2010 Sep 14;122(11):1056-67. doi: 10.1161/CIRCULATIONAHA.109.933796. Epub 2010 Aug 30. PMID 20805430
- [Derived] Cannon CP, Harrington RA, James S, Ardissino D, Becker RC, Emanuelsson H, Husted S, Katus H, Keltai M, Khurmi NS, Kontny F, Lewis BS, Steg PG, Storey RF, Wojdyla D, Wallentin L; PLATelet inhibition and patient Outcomes Investigators. Comparison of ticagrelor with clopidogrel in patients with a planned invasive strategy for acute coronary syndromes (PLATO): a randomised double-blind study. Lancet. 2010 Jan 23;375(9711):283-93. doi: 10.1016/S0140-6736(09)62191-7. Epub 2010 Jan 13. PMID 20079528
- [Derived] Wallentin L, Becker RC, Budaj A, Cannon CP, Emanuelsson H, Held C, Horrow J, Husted S, James S, Katus H, Mahaffey KW, Scirica BM, Skene A, Steg PG, Storey RF, Harrington RA; PLATO Investigators; Freij A, Thorsen M. Ticagrelor versus clopidogrel in patients with acute coronary syndromes. N Engl J Med. 2009 Sep 10;361(11):1045-57. doi: 10.1056/NEJMoa0904327. Epub 2009 Aug 30. PMID 19717846
- [Derived] Molecule of the month. Ticagrelor. Drug News Perspect. 2007 May;20(4):264. No abstract available. PMID 17637939

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first participant was enrolled on 11 October 2006 and the last participant completed the study on 27 February 2009. Study participants were randomized from 855 centers in 43 countries.
Pre-assignment Details: Participants will already be hospitalized due to their acute condition, and must be enrolled and randomized within 24 hours of the onset of their most recent cardiac ischemic symptoms. Randomization should take place as soon as possible after presentation.
Groups:
- TICAGRELOR: Ticagrelor 90 mg twice daily dose (BD)
Period: Overall Study
Arm/Group | TICAGRELOR | CLOPIDOGREL
Started | 9333 | 9291
Completed | 9026 | 9036
Not Completed | 307 | 255
Not completed — Protocol Violation | 7 | 2
Not completed — Withdrawal by Subject | 296 | 249
Not completed — Reason unknown | 2 | 4
Not completed — Lost to Follow-up | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TICAGRELOR | CLOPIDOGREL | Total
Number analyzed (Participants) | 9333 | 9291 | 18624
Age Continuous [Mean (Standard Deviation); unit: years] | 62.1 (11.21) | 62.3 (11.21) | 62.2 (22.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2655 | 2633 | 5288
  Male | 6678 | 6658 | 13336

OUTCOME MEASURES:

1. Primary Outcome: Participants With Any Event From the Composite of Death From Vascular Causes, Myocardial Infarction (MI), and Stroke
Description: Participants with death from vascular causes, MI, or stroke. If no event, censoring occurs at the earliest of patient withdrawal consent or date of scheduled withdrawal from therapy. Intention To Treat (ITT) analysis of whole population. Events were adjudicated by an endpoint committee.
Time Frame: Randomization up to 12 months
Population: The population was the full analysis set, which included all randomized patients
Measure: Number; unit: Participants
Arm/Group | TICAGRELOR | CLOPIDOGREL
Number analyzed (Participants) | 9333 | 9291
Participants | 864 | 1014

2. Primary Outcome: Participants With Any Major Bleeding Event
Description: Participants with major (fatal/life-threatening or other) bleed by a study protocol scale based on need for treatment, number of transfusions, hemoglobin decrease, and other factors. Events were adjudicated by an endpoint committee.
Time Frame: First dosing up to 12 months
Population: The population was the safety analysis set, which included all randomized patients who took at least one dose of study drug
Measure: Number; unit: Participants
Arm/Group | TICAGRELOR | CLOPIDOGREL
Number analyzed (Participants) | 9235 | 9186
Participants | 961 | 929

3. Secondary Outcome: Participants With Any Event From the Composite of Death From Vascular Causes, MI, and Stroke for the Subgroup of Patients With Intent for Invasive Management at Randomization
Description: Participants with death from vascular causes, MI, or stroke. If no event, censoring occurs at the earliest of patient withdrawal consent or date of scheduled withdrawal from therapy. ITT analysis of intent for invasive management population. Events were adjudicated by an endpoint committee.
Time Frame: Randomization up to 12 months
Population: The subgroup of patients with intent for invasive management at randomization
Measure: Number; unit: Participants
Arm/Group | TICAGRELOR | CLOPIDOGREL
Number analyzed (Participants) | 6732 | 6676
Participants | 569 | 668

4. Secondary Outcome: Participants With Any Event From the Composite of All-cause Mortality, MI, and Stroke
Description: Participants with death from any cause, MI, or stroke. If no event, censoring occurs at the earliest of patient withdrawal of consent or date of scheduled withdrawal from therapy. ITT analysis of whole population. Events were adjudicated by an endpoint committee.
Time Frame: Randomization up to 12 months
Population: The population was the full analysis set, which included all randomized patients
Measure: Number; unit: Participants
Arm/Group | TICAGRELOR | CLOPIDOGREL
Number analyzed (Participants) | 9333 | 9291
Participants | 901 | 1065

5. Secondary Outcome: Participants With Any Event From the Composite of Death From Vascular Causes, MI (Including Silent), Stroke, Recurrent Ischemia, Transient Ischemic Attack (TIA) and Other Arterial Thrombotic Events.
Description: Participants with death from vascular causes, MI, stroke, recurrent ischemia, or other thrombotic events. If no event, censoring occurs at the earliest of patient withdrawal consent or date of scheduled withdrawal from therapy. ITT analysis of whole population. Events were adjudicated.
Time Frame: Randomization up to 12 months
Population: The population was the full analysis set, which included all randomized patients
Measure: Number; unit: Participants
Arm/Group | TICAGRELOR | CLOPIDOGREL
Number analyzed (Participants) | 9333 | 9291
Participants | 1290 | 1456

6. Secondary Outcome: Participants With MI Event
Description: Participants with MI event. If no event, censoring occurs at the earliest of patient withdrawal consent or date of scheduled withdrawal from therapy. ITT (intention to treat) analysis of whole population. Events were adjudicated by an endpoint committee.
Time Frame: Randomization up to 12 months
Population: The population was the full analysis set, which included all randomized patients
Measure: Number; unit: Participants
Arm/Group | TICAGRELOR | CLOPIDOGREL
Number analyzed (Participants) | 9333 | 9291
Participants | 504 | 593

7. Secondary Outcome: Participants With Death From Vascular Causes
Description: Participants with death from vascular causes. If no event, censoring occurs at the earliest of patient withdrawal consent or date of scheduled withdrawal from therapy. ITT (intention to treat) analysis of whole population. Events were adjudicated by an endpoint committee.
Time Frame: Randomization up to 12 months
Population: The population was the full analysis set, which included all randomized patients
Measure: Number; unit: Participants
Arm/Group | TICAGRELOR | CLOPIDOGREL
Number analyzed (Participants) | 9333 | 9291
Participants | 353 | 442

8. Secondary Outcome: Participants With Stroke
Description: Participants with stroke. If no event, censoring occurs at the earliest of patient withdrawal consent or date of scheduled withdrawal from therapy. ITT (intention to treat) analysis of whole population. Events were adjudicated by an endpoint committee.
Time Frame: Randomization up to 12 months
Population: The population was the full analysis set, which included all randomized patients
Measure: Number; unit: Participants
Arm/Group | TICAGRELOR | CLOPIDOGREL
Number analyzed (Participants) | 9333 | 9291
Participants | 125 | 106

9. Secondary Outcome: Participants With Death From Any Cause
Description: Participants with death from any cause. If no event, censoring occurs at the earliest of patient withdrawal consent or date of scheduled withdrawal from therapy. ITT (intention to treat) analysis of whole population. Events were adjudicated by an endpoint committee.
Time Frame: Randomization up to 12 months
Population: The population was the full analysis set, which included all randomized patients
Measure: Number; unit: Participants
Arm/Group | TICAGRELOR | CLOPIDOGREL
Number analyzed (Participants) | 9333 | 9291
Participants | 399 | 506

10. Secondary Outcome: Participants With Non-CABG (Coronary Artery Bypass Graft) Related Major Bleeding
Description: Participants with non CABG related major (fatal/life-threatening or other) bleed by a study protocol scale based on need for treatment, number of transfusions, hemoglobin decrease, and other factors. Events were adjudicated by an endpoint committee.
Time Frame: First dosing up to 12 months
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | TICAGRELOR | CLOPIDOGREL
Number analyzed (Participants) | 9235 | 9186
Participants | 362 | 306

11. Secondary Outcome: Participants With Major or Minor Bleeding
Description: Participants with major (fatal/life-threatening or other) or minor bleed by a study protocol scale based on need for treatment, number of transfusions, hemoglobin decrease, and other factors. Events were adjudicated by an endpoint committee.
Time Frame: First dosing up to 12 months
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | TICAGRELOR | CLOPIDOGREL
Number analyzed (Participants) | 9235 | 9186
Participants | 1339 | 1215

12. Secondary Outcome: Participants With Non-procedural Major Bleeding
Description: Participants with non-procedural major bleed by a study protocol scale based on need for treatment, number of transfusions, hemoglobin decrease, and other factors. Events were adjudicated by an endpoint committee.
Time Frame: First dosing up to 12 months
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | TICAGRELOR | CLOPIDOGREL
Number analyzed (Participants) | 9235 | 9186
Participants | 235 | 180

13. Secondary Outcome: Participants With Coronary Artery Bypass Graft (CABG) Major Bleeding
Description: Participants with a major CABG-related bleed by a study protocol scale based on need for treatment, number of transfusions, hemoglobin decrease, and other factors. All CABG surgeries were submitted for adjudication by an endpoint committee as potential bleeds.
Time Frame: First dosing up to 12 months
Population: Population is all patients who underwent CABG surgery within 7 days of last dose of active study medication.
Measure: Number; unit: Participants
Arm/Group | TICAGRELOR | CLOPIDOGREL
Number analyzed (Participants) | 770 | 814
Participants | 619 | 654

14. Secondary Outcome: Participants With Coronary Artery Bypass Graft (CABG) Major Fatal/Life-threatening Bleeding
Description: Number of participants with a major fatal/life-threatening CABG-related bleed by a study protocol scale based on need for treatment, number of transfusions, hemoglobin decrease, and other factors. All CABG surgeries were submitted for adjudication by an endpoint committee as potential bleeds.
Time Frame: First dosing up to 12 months
Population: Population is all patients who underwent CABG surgery within 7 days of last dose of active study medication.
Measure: Number; unit: Participants
Arm/Group | TICAGRELOR | CLOPIDOGREL
Number analyzed (Participants) | 770 | 814
Participants | 329 | 341

15. Secondary Outcome: Participants With Ventricular Pauses of Greater Than or Equal to 3 Seconds in Patients Monitored by Holter 24-hour ECG Recorders for 1 Week Following Randomization
Description: Number of participants who were observed to have at least 1 ventricular pause of at least 3 seconds. Population is all patients who were observed over 2 week-long periods. Pauses were flagged algorithmically and confirmed by Thrombolysis in Myocardial Infarction (TIMI) group cardiologists.
Time Frame: 1-week period following randomization
Population: Participants with Holter data in the week after Randomization
Measure: Number; unit: Participants
Arm/Group | TICAGRELOR | CLOPIDOGREL
Number analyzed (Participants) | 1451 | 1415
Participants | 84 | 51

16. Secondary Outcome: Participants With Ventricular Pauses of Greater Than or Equal to 3 Seconds in Patients Monitored by Holter 24 Hour ECG Recorders for 1 Week at 1 Month Following Randomization
Description: Number of participants who were observed to have at least 1 ventricular pause of at least 3 seconds. Population is all patients who were observed over 2 week-long periods. Pauses were flagged algorithmically and confirmed by TIMI cardiologists.
Time Frame: 1-week period following randomization
Population: Patients who were monitored for one week following randomization (and for one week one month later).
Measure: Number; unit: Participants
Arm/Group | TICAGRELOR | CLOPIDOGREL
Number analyzed (Participants) | 964 | 985
Participants | 21 | 16

ADVERSE EVENTS:
Arm/Group | TICAGRELOR | CLOPIDOGREL
Serious Adverse Events (participants affected / at risk) | 2108 | 2117
Other Adverse Events (participants affected / at risk) | 2278 | 1665
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | TICAGRELOR | CLOPIDOGREL
Anaemia (Blood and lymphatic system disorders) | 35/9333 | 25/9291
Thrombocytopenia (Blood and lymphatic system disorders) | 7/9333 | 8/9291
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 2/9333 | 6/9291
Leukopenia (Blood and lymphatic system disorders) | 1/9333 | 2/9291
Lymphadenitis (Blood and lymphatic system disorders) | 2/9333 | 0/9291
Microcytic Anaemia (Blood and lymphatic system disorders) | 1/9333 | 2/9291
Spontaneous Haematoma (Blood and lymphatic system disorders) | 2/9333 | 0/9291
Coagulopathy (Blood and lymphatic system disorders) | 1/9333 | 0/9291
Disseminated Intravascular Coagulation (Blood and lymphatic system disorders) | 0/9333 | 1/9291
Granulocytopenia (Blood and lymphatic system disorders) | 1/9333 | 0/9291
Haemorrhagic Anaemia (Blood and lymphatic system disorders) | 1/9333 | 0/9291
Hypochromic Anaemia (Blood and lymphatic system disorders) | 1/9333 | 0/9291
Leukocytosis (Blood and lymphatic system disorders) | 0/9333 | 1/9291
Lymphadenopathy (Blood and lymphatic system disorders) | 0/9333 | 1/9291
Nephrogenic Anaemia (Blood and lymphatic system disorders) | 1/9333 | 0/9291
Neutropenia (Blood and lymphatic system disorders) | 1/9333 | 1/9291
Normochromic Normocytic Anaemia (Blood and lymphatic system disorders) | 1/9333 | 0/9291
Pancytopenia (Blood and lymphatic system disorders) | 1/9333 | 0/9291
Polycythaemia (Blood and lymphatic system disorders) | 1/9333 | 1/9291
Splenic Lesion (Blood and lymphatic system disorders) | 1/9333 | 0/9291
Thrombocythaemia (Blood and lymphatic system disorders) | 0/9333 | 1/9291
Cardiac Failure (Cardiac disorders) | 122/9333 | 129/9291
Atrial Fibrillation (Cardiac disorders) | 70/9333 | 68/9291
Cardiogenic Shock (Cardiac disorders) | 60/9333 | 66/9291
Ventricular Fibrillation (Cardiac disorders) | 48/9333 | 64/9291
Cardiac Failure Congestive (Cardiac disorders) | 51/9333 | 46/9291
Cardiac Arrest (Cardiac disorders) | 38/9333 | 44/9291
Ventricular Tachycardia (Cardiac disorders) | 29/9333 | 33/9291
Bradycardia (Cardiac disorders) | 26/9333 | 31/9291
Atrioventricular Block Complete (Cardiac disorders) | 19/9333 | 19/9291
Cardiac Failure Acute (Cardiac disorders) | 18/9333 | 18/9291
Cardiac Tamponade (Cardiac disorders) | 11/9333 | 16/9291
Intracardiac Thrombus (Cardiac disorders) | 13/9333 | 15/9291
Angina Pectoris (Cardiac disorders) | 7/9333 | 14/9291
Cardio-Respiratory Arrest (Cardiac disorders) | 8/9333 | 12/9291
Atrial Flutter (Cardiac disorders) | 11/9333 | 7/9291
Left Ventricular Failure (Cardiac disorders) | 10/9333 | 5/9291
Pericardial Effusion (Cardiac disorders) | 9/9333 | 10/9291
Arrhythmia (Cardiac disorders) | 8/9333 | 4/9291
Palpitations (Cardiac disorders) | 8/9333 | 7/9291
Pericarditis (Cardiac disorders) | 6/9333 | 8/9291
Supraventricular Tachycardia (Cardiac disorders) | 8/9333 | 8/9291
Sick Sinus Syndrome (Cardiac disorders) | 7/9333 | 2/9291
Cardiac Asthma (Cardiac disorders) | 3/9333 | 6/9291
Mitral Valve Incompetence (Cardiac disorders) | 4/9333 | 6/9291
Ventricular Arrhythmia (Cardiac disorders) | 3/9333 | 6/9291
Ventricular Extrasystoles (Cardiac disorders) | 6/9333 | 1/9291
Atrioventricular Block (Cardiac disorders) | 3/9333 | 5/9291
Cardiac Failure Chronic (Cardiac disorders) | 5/9333 | 2/9291
Coronary Artery Disease (Cardiac disorders) | 5/9333 | 3/9291
Coronary Artery Dissection (Cardiac disorders) | 5/9333 | 3/9291
Atrioventricular Block Second Degree (Cardiac disorders) | 4/9333 | 0/9291
Electromechanical Dissociation (Cardiac disorders) | 3/9333 | 4/9291
Myocardial Rupture (Cardiac disorders) | 2/9333 | 4/9291
Sinus Bradycardia (Cardiac disorders) | 1/9333 | 4/9291
Tachyarrhythmia (Cardiac disorders) | 4/9333 | 4/9291
Tachycardia (Cardiac disorders) | 1/9333 | 4/9291
Acute Left Ventricular Failure (Cardiac disorders) | 3/9333 | 2/9291
Aortic Valve Stenosis (Cardiac disorders) | 2/9333 | 3/9291
Atrial Tachycardia (Cardiac disorders) | 1/9333 | 3/9291
Bradyarrhythmia (Cardiac disorders) | 3/9333 | 3/9291
Cardiac Aneurysm (Cardiac disorders) | 1/9333 | 3/9291
Cardiomyopathy (Cardiac disorders) | 1/9333 | 3/9291
Coronary Artery Perforation (Cardiac disorders) | 3/9333 | 0/9291
Coronary Artery Thrombosis (Cardiac disorders) | 2/9333 | 3/9291
Dressler's Syndrome (Cardiac disorders) | 3/9333 | 3/9291
Left Ventricular Dysfunction (Cardiac disorders) | 3/9333 | 3/9291
Pericardial Haemorrhage (Cardiac disorders) | 3/9333 | 2/9291
Sinus Arrest (Cardiac disorders) | 1/9333 | 3/9291
Ventricle Rupture (Cardiac disorders) | 2/9333 | 3/9291
Arrhythmia Supraventricular (Cardiac disorders) | 1/9333 | 2/9291
Arteriosclerosis Coronary Artery (Cardiac disorders) | 0/9333 | 2/9291
Cardiopulmonary Failure (Cardiac disorders) | 1/9333 | 2/9291
Coronary Artery Occlusion (Cardiac disorders) | 0/9333 | 2/9291
Coronary Artery Stenosis (Cardiac disorders) | 2/9333 | 1/9291
Nodal Rhythm (Cardiac disorders) | 1/9333 | 2/9291
Papillary Muscle Rupture (Cardiac disorders) | 2/9333 | 1/9291
Right Ventricular Failure (Cardiac disorders) | 2/9333 | 1/9291
Acute Coronary Syndrome (Cardiac disorders) | 1/9333 | 1/9291
Arteriospasm Coronary (Cardiac disorders) | 1/9333 | 0/9291
Atrial Rupture (Cardiac disorders) | 1/9333 | 0/9291
Bundle Branch Block (Cardiac disorders) | 0/9333 | 1/9291
Bundle Branch Block Left (Cardiac disorders) | 0/9333 | 1/9291
Cardiac Disorder (Cardiac disorders) | 0/9333 | 1/9291
Cardiac Valve Disease (Cardiac disorders) | 1/9333 | 0/9291
Cardiovascular Disorder (Cardiac disorders) | 0/9333 | 1/9291
Chordae Tendinae Rupture (Cardiac disorders) | 0/9333 | 1/9291
Coronary Artery Insufficiency (Cardiac disorders) | 0/9333 | 1/9291
Cyanosis (Cardiac disorders) | 1/9333 | 0/9291
Dissecting Coronary Artery Aneurysm (Cardiac disorders) | 0/9333 | 1/9291
Extrasystoles (Cardiac disorders) | 1/9333 | 1/9291
Hypertrophic Cardiomyopathy (Cardiac disorders) | 1/9333 | 1/9291
Interventricular Septum Rupture (Cardiac disorders) | 1/9333 | 0/9291
Ischaemic Cardiomyopathy (Cardiac disorders) | 1/9333 | 0/9291
Long Qt Syndrome (Cardiac disorders) | 0/9333 | 1/9291
Low Cardiac Output Syndrome (Cardiac disorders) | 0/9333 | 1/9291
Myocardial Infarction (Cardiac disorders) | 0/9333 | 1/9291
Myocardial Ischaemia (Cardiac disorders) | 0/9333 | 1/9291
Myocarditis (Cardiac disorders) | 1/9333 | 0/9291
Papillary Muscle Disorder (Cardiac disorders) | 0/9333 | 1/9291
Stress Cardiomyopathy (Cardiac disorders) | 0/9333 | 1/9291
Torsade De Pointes (Cardiac disorders) | 0/9333 | 1/9291
Ventricular Dysfunction (Cardiac disorders) | 0/9333 | 1/9291
Ventricular Tachyarrhythmia (Cardiac disorders) | 0/9333 | 1/9291
Carbohydrate Metabolism Disorder (Congenital, familial and genetic disorders) | 0/9333 | 2/9291
Diverticulitis Meckel's (Congenital, familial and genetic disorders) | 1/9333 | 0/9291
Gastrointestinal Angiodysplasia Haemorrhagic (Congenital, familial and genetic disorders) | 0/9333 | 1/9291
Haemorrhagic Arteriovenous Malformation (Congenital, familial and genetic disorders) | 1/9333 | 0/9291
Ventricular Septal Defect (Congenital, familial and genetic disorders) | 0/9333 | 1/9291
Vertigo (Ear and labyrinth disorders) | 8/9333 | 5/9291
Vestibular Neuronitis (Ear and labyrinth disorders) | 1/9333 | 3/9291
Hypoacusis (Ear and labyrinth disorders) | 2/9333 | 0/9291
Deafness (Ear and labyrinth disorders) | 1/9333 | 0/9291
Sudden Hearing Loss (Ear and labyrinth disorders) | 0/9333 | 1/9291
Tinnitus (Ear and labyrinth disorders) | 1/9333 | 0/9291
Vertigo Positional (Ear and labyrinth disorders) | 1/9333 | 0/9291
Hyperthyroidism (Endocrine disorders) | 2/9333 | 2/9291
Goitre (Endocrine disorders) | 0/9333 | 1/9291
Pituitary-Dependent Cushing's Syndrome (Endocrine disorders) | 1/9333 | 0/9291
Thyrotoxic Crisis (Endocrine disorders) | 0/9333 | 1/9291
Cataract (Eye disorders) | 3/9333 | 2/9291
Diplopia (Eye disorders) | 2/9333 | 1/9291
Retinal Detachment (Eye disorders) | 2/9333 | 2/9291
Amaurosis (Eye disorders) | 1/9333 | 0/9291
Amaurosis Fugax (Eye disorders) | 0/9333 | 1/9291
Blindness (Eye disorders) | 1/9333 | 0/9291
Cataract Nuclear (Eye disorders) | 1/9333 | 0/9291
Chorioretinitis (Eye disorders) | 0/9333 | 1/9291
Conjunctival Haemorrhage (Eye disorders) | 1/9333 | 0/9291
Diabetic Retinopathy (Eye disorders) | 1/9333 | 0/9291
Eye Haemorrhage (Eye disorders) | 1/9333 | 1/9291
Glaucoma (Eye disorders) | 1/9333 | 0/9291
Macular Degeneration (Eye disorders) | 1/9333 | 1/9291
Posterior Capsule Opacification (Eye disorders) | 0/9333 | 1/9291
Retinal Artery Embolism (Eye disorders) | 0/9333 | 1/9291
Visual Impairment (Eye disorders) | 1/9333 | 1/9291
Vitreous Haemorrhage (Eye disorders) | 1/9333 | 0/9291
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 45/9333 | 42/9291
Abdominal Pain (Gastrointestinal disorders) | 21/9333 | 10/9291
Abdominal Pain Upper (Gastrointestinal disorders) | 9/9333 | 15/9291
Diarrhoea (Gastrointestinal disorders) | 12/9333 | 9/9291
Gastric Ulcer Haemorrhage (Gastrointestinal disorders) | 11/9333 | 6/9291
Duodenal Ulcer Haemorrhage (Gastrointestinal disorders) | 10/9333 | 2/9291
Melaena (Gastrointestinal disorders) | 10/9333 | 3/9291
Vomiting (Gastrointestinal disorders) | 10/9333 | 4/9291
Gastritis (Gastrointestinal disorders) | 8/9333 | 9/9291
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 9/9333 | 7/9291
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 4/9333 | 7/9291
Rectal Haemorrhage (Gastrointestinal disorders) | 7/9333 | 6/9291
Dyspepsia (Gastrointestinal disorders) | 6/9333 | 5/9291
Haematemesis (Gastrointestinal disorders) | 5/9333 | 3/9291
Pancreatitis (Gastrointestinal disorders) | 4/9333 | 5/9291
Pancreatitis Acute (Gastrointestinal disorders) | 5/9333 | 1/9291
Retroperitoneal Haemorrhage (Gastrointestinal disorders) | 5/9333 | 3/9291
Gastric Haemorrhage (Gastrointestinal disorders) | 3/9333 | 4/9291
Gastric Ulcer (Gastrointestinal disorders) | 4/9333 | 2/9291
Gastritis Erosive (Gastrointestinal disorders) | 4/9333 | 2/9291
Haematochezia (Gastrointestinal disorders) | 4/9333 | 2/9291
Inguinal Hernia (Gastrointestinal disorders) | 4/9333 | 4/9291
Lower Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1/9333 | 4/9291
Nausea (Gastrointestinal disorders) | 3/9333 | 4/9291
Anal Haemorrhage (Gastrointestinal disorders) | 0/9333 | 3/9291
Diverticulum (Gastrointestinal disorders) | 3/9333 | 0/9291
Duodenal Ulcer (Gastrointestinal disorders) | 3/9333 | 2/9291
Enteritis (Gastrointestinal disorders) | 0/9333 | 3/9291
Gastrointestinal Necrosis (Gastrointestinal disorders) | 3/9333 | 0/9291
Haemorrhoidal Haemorrhage (Gastrointestinal disorders) | 2/9333 | 3/9291
Peptic Ulcer Haemorrhage (Gastrointestinal disorders) | 3/9333 | 1/9291
Peritonitis (Gastrointestinal disorders) | 1/9333 | 3/9291
Retroperitoneal Haematoma (Gastrointestinal disorders) | 3/9333 | 3/9291
Abdominal Discomfort (Gastrointestinal disorders) | 0/9333 | 2/9291
Constipation (Gastrointestinal disorders) | 1/9333 | 2/9291
Diverticulum Intestinal (Gastrointestinal disorders) | 2/9333 | 0/9291
Diverticulum Intestinal Haemorrhagic (Gastrointestinal disorders) | 1/9333 | 2/9291
Duodenitis (Gastrointestinal disorders) | 0/9333 | 2/9291
Dysphagia (Gastrointestinal disorders) | 2/9333 | 2/9291
Faeces Discoloured (Gastrointestinal disorders) | 2/9333 | 0/9291
Gastric Disorder (Gastrointestinal disorders) | 0/9333 | 2/9291
Gastritis Haemorrhagic (Gastrointestinal disorders) | 1/9333 | 2/9291
Gastroduodenal Haemorrhage (Gastrointestinal disorders) | 2/9333 | 0/9291
Ileus Paralytic (Gastrointestinal disorders) | 2/9333 | 0/9291
Intestinal Haemorrhage (Gastrointestinal disorders) | 1/9333 | 2/9291
Intestinal Ischaemia (Gastrointestinal disorders) | 0/9333 | 2/9291
Large Intestine Perforation (Gastrointestinal disorders) | 2/9333 | 1/9291
Oesophagitis (Gastrointestinal disorders) | 1/9333 | 2/9291
Rectal Polyp (Gastrointestinal disorders) | 2/9333 | 0/9291
Small Intestinal Obstruction (Gastrointestinal disorders) | 2/9333 | 1/9291
Abdominal Hernia Obstructive (Gastrointestinal disorders) | 1/9333 | 0/9291
Anal Fistula (Gastrointestinal disorders) | 0/9333 | 1/9291
Appendicitis Perforated (Gastrointestinal disorders) | 1/9333 | 0/9291
Ascites (Gastrointestinal disorders) | 0/9333 | 1/9291
Colitis Ischaemic (Gastrointestinal disorders) | 0/9333 | 1/9291
Colitis Ulcerative (Gastrointestinal disorders) | 0/9333 | 1/9291
Colonic Polyp (Gastrointestinal disorders) | 1/9333 | 1/9291
Dental Caries (Gastrointestinal disorders) | 0/9333 | 1/9291
Diarrhoea Haemorrhagic (Gastrointestinal disorders) | 1/9333 | 0/9291
Diverticular Perforation (Gastrointestinal disorders) | 0/9333 | 1/9291
Diverticulitis Intestinal Haemorrhagic (Gastrointestinal disorders) | 1/9333 | 0/9291
Enterocolitis Haemorrhagic (Gastrointestinal disorders) | 1/9333 | 0/9291
Epigastric Discomfort (Gastrointestinal disorders) | 1/9333 | 0/9291
Erosive Oesophagitis (Gastrointestinal disorders) | 1/9333 | 0/9291
Faecal Incontinence (Gastrointestinal disorders) | 0/9333 | 1/9291
Food Poisoning (Gastrointestinal disorders) | 0/9333 | 1/9291
Gastritis Atrophic (Gastrointestinal disorders) | 0/9333 | 1/9291
Gastrointestinal Disorder (Gastrointestinal disorders) | 1/9333 | 1/9291
Gastrointestinal Pain (Gastrointestinal disorders) | 1/9333 | 0/9291
Gastrointestinal Ulcer Haemorrhage (Gastrointestinal disorders) | 1/9333 | 0/9291
Gingival Bleeding (Gastrointestinal disorders) | 1/9333 | 0/9291
Gingivitis Ulcerative (Gastrointestinal disorders) | 0/9333 | 1/9291
Haemorrhagic Erosive Gastritis (Gastrointestinal disorders) | 0/9333 | 1/9291
Haemorrhoids (Gastrointestinal disorders) | 1/9333 | 1/9291
Hiatus Hernia (Gastrointestinal disorders) | 0/9333 | 1/9291
Inguinal Hernia Strangulated (Gastrointestinal disorders) | 0/9333 | 1/9291
Intestinal Obstruction (Gastrointestinal disorders) | 0/9333 | 1/9291
Intestinal Polyp (Gastrointestinal disorders) | 1/9333 | 0/9291
Intra-Abdominal Haemorrhage (Gastrointestinal disorders) | 1/9333 | 1/9291
Mallory-Weiss Syndrome (Gastrointestinal disorders) | 0/9333 | 1/9291
Mesenteric Artery Embolism (Gastrointestinal disorders) | 0/9333 | 1/9291
Mouth Haemorrhage (Gastrointestinal disorders) | 0/9333 | 1/9291
Oesophageal Food Impaction (Gastrointestinal disorders) | 1/9333 | 0/9291
Oesophageal Haemorrhage (Gastrointestinal disorders) | 0/9333 | 1/9291
Oesophageal Pain (Gastrointestinal disorders) | 1/9333 | 0/9291
Oesophageal Varices Haemorrhage (Gastrointestinal disorders) | 0/9333 | 1/9291
Oesophagitis Haemorrhagic (Gastrointestinal disorders) | 1/9333 | 0/9291
Pancreatic Disorder (Gastrointestinal disorders) | 0/9333 | 1/9291
Pancreatic Haemorrhage (Gastrointestinal disorders) | 0/9333 | 1/9291
Pancreatitis Chronic (Gastrointestinal disorders) | 1/9333 | 0/9291
Peptic Ulcer (Gastrointestinal disorders) | 0/9333 | 1/9291
Pneumoperitoneum (Gastrointestinal disorders) | 1/9333 | 0/9291
Polyp Colorectal (Gastrointestinal disorders) | 0/9333 | 1/9291
Proctitis (Gastrointestinal disorders) | 1/9333 | 0/9291
Reflux Oesophagitis (Gastrointestinal disorders) | 1/9333 | 0/9291
Retroperitoneal Fibrosis (Gastrointestinal disorders) | 1/9333 | 0/9291
Small Intestinal Haemorrhage (Gastrointestinal disorders) | 1/9333 | 0/9291
Small Intestinal Perforation (Gastrointestinal disorders) | 1/9333 | 0/9291
Stomach Mass (Gastrointestinal disorders) | 1/9333 | 0/9291
Subileus (Gastrointestinal disorders) | 1/9333 | 0/9291
Thrombosis Mesenteric Vessel (Gastrointestinal disorders) | 0/9333 | 1/9291
Tongue Oedema (Gastrointestinal disorders) | 1/9333 | 0/9291
Toothache (Gastrointestinal disorders) | 1/9333 | 0/9291
Volvulus (Gastrointestinal disorders) | 0/9333 | 1/9291
Non-Cardiac Chest Pain (General disorders) | 101/9333 | 103/9291
Chest Pain (General disorders) | 54/9333 | 63/9291
Death (General disorders) | 21/9333 | 31/9291
Sudden Death (General disorders) | 17/9333 | 27/9291
Sudden Cardiac Death (General disorders) | 14/9333 | 25/9291
Vessel Puncture Site Haematoma (General disorders) | 8/9333 | 12/9291
Pyrexia (General disorders) | 10/9333 | 5/9291
Multi-Organ Failure (General disorders) | 9/9333 | 9/9291
Vessel Puncture Site Haemorrhage (General disorders) | 9/9333 | 6/9291
Asthenia (General disorders) | 6/9333 | 4/9291
Malaise (General disorders) | 6/9333 | 3/9291
General Physical Health Deterioration (General disorders) | 1/9333 | 5/9291
Chest Discomfort (General disorders) | 4/9333 | 2/9291
Impaired Healing (General disorders) | 1/9333 | 4/9291
Oedema Peripheral (General disorders) | 4/9333 | 1/9291
Puncture Site Haemorrhage (General disorders) | 4/9333 | 1/9291
Cardiac Death (General disorders) | 3/9333 | 1/9291
Catheter Site Haemorrhage (General disorders) | 1/9333 | 2/9291
Fatigue (General disorders) | 1/9333 | 2/9291
Systemic Inflammatory Response Syndrome (General disorders) | 1/9333 | 2/9291
Accidental Death (General disorders) | 1/9333 | 0/9291
Alcohol Interaction (General disorders) | 1/9333 | 0/9291
Application Site Inflammation (General disorders) | 1/9333 | 0/9291
Discomfort (General disorders) | 1/9333 | 0/9291
Foaming At Mouth (General disorders) | 1/9333 | 0/9291
Gait Disturbance (General disorders) | 0/9333 | 1/9291
Generalised Oedema (General disorders) | 1/9333 | 0/9291
Hernia (General disorders) | 1/9333 | 0/9291
Hypothermia (General disorders) | 1/9333 | 0/9291
Inflammation (General disorders) | 0/9333 | 1/9291
Inflammation Of Wound (General disorders) | 1/9333 | 0/9291
Injection Site Haemorrhage (General disorders) | 1/9333 | 0/9291
Injection Site Swelling (General disorders) | 1/9333 | 0/9291
Pain (General disorders) | 0/9333 | 1/9291
Pelvic Mass (General disorders) | 0/9333 | 1/9291
Ulcer Haemorrhage (General disorders) | 1/9333 | 1/9291
Unevaluable Event (General disorders) | 1/9333 | 0/9291
Cholecystitis (Hepatobiliary disorders) | 7/9333 | 10/9291
Cholelithiasis (Hepatobiliary disorders) | 9/9333 | 9/9291
Cholecystitis Acute (Hepatobiliary disorders) | 5/9333 | 7/9291
Hepatic Failure (Hepatobiliary disorders) | 2/9333 | 4/9291
Bile Duct Stone (Hepatobiliary disorders) | 2/9333 | 2/9291
Biliary Colic (Hepatobiliary disorders) | 1/9333 | 2/9291
Cholangitis (Hepatobiliary disorders) | 1/9333 | 2/9291
Hepatic Cirrhosis (Hepatobiliary disorders) | 1/9333 | 2/9291
Jaundice (Hepatobiliary disorders) | 0/9333 | 2/9291
Bile Duct Obstruction (Hepatobiliary disorders) | 1/9333 | 0/9291
Cholecystitis Chronic (Hepatobiliary disorders) | 1/9333 | 0/9291
Cholestasis (Hepatobiliary disorders) | 1/9333 | 0/9291
Gallbladder Disorder (Hepatobiliary disorders) | 1/9333 | 0/9291
Gallbladder Necrosis (Hepatobiliary disorders) | 1/9333 | 0/9291
Hepatic Function Abnormal (Hepatobiliary disorders) | 1/9333 | 0/9291
Hepatitis Toxic (Hepatobiliary disorders) | 1/9333 | 0/9291
Hepatocellular Injury (Hepatobiliary disorders) | 1/9333 | 0/9291
Ischaemic Hepatitis (Hepatobiliary disorders) | 1/9333 | 0/9291
Liver Disorder (Hepatobiliary disorders) | 1/9333 | 0/9291
Anaphylactic Reaction (Immune system disorders) | 0/9333 | 3/9291
Anaphylactic Shock (Immune system disorders) | 3/9333 | 1/9291
Drug Hypersensitivity (Immune system disorders) | 1/9333 | 3/9291
Hypersensitivity (Immune system disorders) | 1/9333 | 2/9291
Allergy To Arthropod Bite (Immune system disorders) | 0/9333 | 1/9291
Contrast Media Allergy (Immune system disorders) | 0/9333 | 1/9291
Pneumonia (Infections and infestations) | 69/9333 | 95/9291
Sepsis (Infections and infestations) | 17/9333 | 27/9291
Urinary Tract Infection (Infections and infestations) | 25/9333 | 19/9291
Gastroenteritis (Infections and infestations) | 17/9333 | 11/9291
Bronchitis (Infections and infestations) | 13/9333 | 15/9291
Mediastinitis (Infections and infestations) | 11/9333 | 4/9291
Bronchopneumonia (Infections and infestations) | 10/9333 | 4/9291
Septic Shock (Infections and infestations) | 5/9333 | 10/9291
Cellulitis (Infections and infestations) | 9/9333 | 9/9291
Postoperative Wound Infection (Infections and infestations) | 9/9333 | 3/9291
Respiratory Tract Infection (Infections and infestations) | 9/9333 | 5/9291
Diverticulitis (Infections and infestations) | 7/9333 | 8/9291
Wound Infection (Infections and infestations) | 7/9333 | 8/9291
Appendicitis (Infections and infestations) | 6/9333 | 2/9291
Infection (Infections and infestations) | 1/9333 | 5/9291
Lung Infection (Infections and infestations) | 5/9333 | 4/9291
Erysipelas (Infections and infestations) | 4/9333 | 4/9291
Lower Respiratory Tract Infection (Infections and infestations) | 3/9333 | 4/9291
Urosepsis (Infections and infestations) | 4/9333 | 2/9291
Cystitis (Infections and infestations) | 3/9333 | 2/9291
Endocarditis (Infections and infestations) | 3/9333 | 2/9291
Gangrene (Infections and infestations) | 2/9333 | 3/9291
Gastrointestinal Infection (Infections and infestations) | 3/9333 | 1/9291
Osteomyelitis (Infections and infestations) | 3/9333 | 3/9291
Pyelonephritis (Infections and infestations) | 3/9333 | 2/9291
Staphylococcal Sepsis (Infections and infestations) | 3/9333 | 1/9291
Upper Respiratory Tract Infection (Infections and infestations) | 3/9333 | 3/9291
Abscess Limb (Infections and infestations) | 2/9333 | 0/9291
Acute Tonsillitis (Infections and infestations) | 2/9333 | 0/9291
Anal Abscess (Infections and infestations) | 2/9333 | 2/9291
Bacteraemia (Infections and infestations) | 2/9333 | 1/9291
Gastroenteritis Caliciviral (Infections and infestations) | 2/9333 | 0/9291
Gastroenteritis Viral (Infections and infestations) | 2/9333 | 0/9291
Incision Site Infection (Infections and infestations) | 2/9333 | 1/9291
Lobar Pneumonia (Infections and infestations) | 0/9333 | 2/9291
Localised Infection (Infections and infestations) | 0/9333 | 2/9291
Sinusitis (Infections and infestations) | 2/9333 | 0/9291
Skin Infection (Infections and infestations) | 2/9333 | 2/9291
Staphylococcal Infection (Infections and infestations) | 2/9333 | 0/9291
Tooth Abscess (Infections and infestations) | 0/9333 | 2/9291
Abdominal Abscess (Infections and infestations) | 1/9333 | 1/9291
Abdominal Wall Infection (Infections and infestations) | 0/9333 | 1/9291
Abscess (Infections and infestations) | 1/9333 | 0/9291
Acquired Immunodeficiency Syndrome (Infections and infestations) | 1/9333 | 0/9291
Acute Sinusitis (Infections and infestations) | 1/9333 | 0/9291
Arthritis Bacterial (Infections and infestations) | 1/9333 | 0/9291
Arthritis Infective (Infections and infestations) | 1/9333 | 1/9291
Bacterial Infection (Infections and infestations) | 1/9333 | 1/9291
Breast Abscess (Infections and infestations) | 0/9333 | 1/9291
Bronchiectasis (Infections and infestations) | 1/9333 | 0/9291
Bronchitis Viral (Infections and infestations) | 0/9333 | 1/9291
Catheter Related Infection (Infections and infestations) | 1/9333 | 0/9291
Catheter Site Infection (Infections and infestations) | 0/9333 | 1/9291
Cholecystitis Infective (Infections and infestations) | 0/9333 | 1/9291
Clostridium Difficile Colitis (Infections and infestations) | 1/9333 | 1/9291
Dengue Fever (Infections and infestations) | 0/9333 | 1/9291
Device Related Infection (Infections and infestations) | 1/9333 | 0/9291
Diarrhoea Infectious (Infections and infestations) | 1/9333 | 0/9291
Endometritis (Infections and infestations) | 1/9333 | 0/9291
Enterococcal Infection (Infections and infestations) | 0/9333 | 1/9291
Enterocolitis Infectious (Infections and infestations) | 1/9333 | 0/9291
Febrile Infection (Infections and infestations) | 1/9333 | 0/9291
Gastric Infection (Infections and infestations) | 1/9333 | 0/9291
Gastroenteritis Rotavirus (Infections and infestations) | 0/9333 | 1/9291
Gastroenteritis Salmonella (Infections and infestations) | 1/9333 | 0/9291
Groin Abscess (Infections and infestations) | 0/9333 | 1/9291
Groin Infection (Infections and infestations) | 1/9333 | 0/9291
Haematoma Infection (Infections and infestations) | 1/9333 | 0/9291
Helicobacter Gastritis (Infections and infestations) | 1/9333 | 1/9291
Hepatitis Viral (Infections and infestations) | 1/9333 | 0/9291
Herpes Zoster (Infections and infestations) | 1/9333 | 1/9291
Histoplasmosis (Infections and infestations) | 1/9333 | 0/9291
Impetigo (Infections and infestations) | 0/9333 | 1/9291
Incision Site Abscess (Infections and infestations) | 1/9333 | 0/9291
Infected Skin Ulcer (Infections and infestations) | 1/9333 | 0/9291
Infective Exacerbation Of Chronic Obstructive Airways Disease (Infections and infestations) | 1/9333 | 0/9291
Infective Tenosynovitis (Infections and infestations) | 0/9333 | 1/9291
Inguinal Hernia Gangrenous (Infections and infestations) | 0/9333 | 1/9291
Injection Site Cellulitis (Infections and infestations) | 0/9333 | 1/9291
Intervertebral Discitis (Infections and infestations) | 0/9333 | 1/9291
Laryngitis (Infections and infestations) | 1/9333 | 0/9291
Liver Abscess (Infections and infestations) | 1/9333 | 0/9291
Lyme Disease (Infections and infestations) | 0/9333 | 1/9291
Meningitis (Infections and infestations) | 0/9333 | 1/9291
Necrotising Fasciitis (Infections and infestations) | 1/9333 | 0/9291
Orchitis (Infections and infestations) | 0/9333 | 1/9291
Pancreatic Abscess (Infections and infestations) | 1/9333 | 0/9291
Perineal Abscess (Infections and infestations) | 1/9333 | 0/9291
Pharyngitis (Infections and infestations) | 0/9333 | 1/9291
Pneumococcal Sepsis (Infections and infestations) | 0/9333 | 1/9291
Pneumonia Staphylococcal (Infections and infestations) | 0/9333 | 1/9291
Post Procedural Cellulitis (Infections and infestations) | 0/9333 | 1/9291
Post Procedural Infection (Infections and infestations) | 1/9333 | 1/9291
Post Procedural Sepsis (Infections and infestations) | 0/9333 | 1/9291
Pulmonary Sepsis (Infections and infestations) | 1/9333 | 0/9291
Pulmonary Tuberculosis (Infections and infestations) | 1/9333 | 0/9291
Puncture Site Abscess (Infections and infestations) | 1/9333 | 0/9291
Puncture Site Infection (Infections and infestations) | 0/9333 | 1/9291
Pyelonephritis Acute (Infections and infestations) | 1/9333 | 1/9291
Pyothorax (Infections and infestations) | 1/9333 | 0/9291
Rectal Abscess (Infections and infestations) | 0/9333 | 1/9291
Renal Abscess (Infections and infestations) | 1/9333 | 1/9291
Retroperitoneal Abscess (Infections and infestations) | 0/9333 | 1/9291
Staphylococcal Mediastinitis (Infections and infestations) | 0/9333 | 1/9291
Sternitis (Infections and infestations) | 1/9333 | 1/9291
Subcutaneous Abscess (Infections and infestations) | 0/9333 | 1/9291
Syphilis (Infections and infestations) | 1/9333 | 0/9291
Tooth Infection (Infections and infestations) | 0/9333 | 1/9291
Tracheitis (Infections and infestations) | 1/9333 | 0/9291
Tracheobronchitis (Infections and infestations) | 1/9333 | 1/9291
Viral Myocarditis (Infections and infestations) | 1/9333 | 1/9291
Viral Pericarditis (Infections and infestations) | 0/9333 | 1/9291
Thrombosis In Device (Injury, poisoning and procedural complications) | 35/9333 | 57/9291
Post Procedural Haemorrhage (Injury, poisoning and procedural complications) | 56/9333 | 47/9291
In-Stent Coronary Artery Restenosis (Injury, poisoning and procedural complications) | 35/9333 | 25/9291
Vascular Pseudoaneurysm (Injury, poisoning and procedural complications) | 15/9333 | 23/9291
In-Stent Arterial Restenosis (Injury, poisoning and procedural complications) | 10/9333 | 12/9291
Coronary Artery Restenosis (Injury, poisoning and procedural complications) | 4/9333 | 9/9291
Femur Fracture (Injury, poisoning and procedural complications) | 3/9333 | 7/9291
Post Procedural Haematoma (Injury, poisoning and procedural complications) | 7/9333 | 1/9291
Fall (Injury, poisoning and procedural complications) | 1/9333 | 5/9291
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 3/9333 | 5/9291
Postpericardiotomy Syndrome (Injury, poisoning and procedural complications) | 5/9333 | 2/9291
Hip Fracture (Injury, poisoning and procedural complications) | 4/9333 | 2/9291
Lower Limb Fracture (Injury, poisoning and procedural complications) | 0/9333 | 4/9291
Post Procedural Complication (Injury, poisoning and procedural complications) | 4/9333 | 4/9291
Subdural Haematoma (Injury, poisoning and procedural complications) | 4/9333 | 2/9291
Wrist Fracture (Injury, poisoning and procedural complications) | 4/9333 | 0/9291
Hand Fracture (Injury, poisoning and procedural complications) | 3/9333 | 0/9291
Head Injury (Injury, poisoning and procedural complications) | 1/9333 | 3/9291
Injury (Injury, poisoning and procedural complications) | 1/9333 | 3/9291
Operative Haemorrhage (Injury, poisoning and procedural complications) | 2/9333 | 3/9291
Postoperative Thoracic Procedure Complication (Injury, poisoning and procedural complications) | 3/9333 | 3/9291
Postoperative Wound Complication (Injury, poisoning and procedural complications) | 2/9333 | 3/9291
Procedural Pain (Injury, poisoning and procedural complications) | 3/9333 | 0/9291
Subcutaneous Haematoma (Injury, poisoning and procedural complications) | 3/9333 | 0/9291
Wound Dehiscence (Injury, poisoning and procedural complications) | 3/9333 | 2/9291
Alcohol Poisoning (Injury, poisoning and procedural complications) | 2/9333 | 0/9291
Clavicle Fracture (Injury, poisoning and procedural complications) | 0/9333 | 2/9291
Concussion (Injury, poisoning and procedural complications) | 2/9333 | 2/9291
Facial Bones Fracture (Injury, poisoning and procedural complications) | 2/9333 | 1/9291
Foot Fracture (Injury, poisoning and procedural complications) | 0/9333 | 2/9291
Graft Thrombosis (Injury, poisoning and procedural complications) | 0/9333 | 2/9291
Humerus Fracture (Injury, poisoning and procedural complications) | 2/9333 | 1/9291
Ligament Rupture (Injury, poisoning and procedural complications) | 2/9333 | 0/9291
Limb Injury (Injury, poisoning and procedural complications) | 2/9333 | 0/9291
Limb Traumatic Amputation (Injury, poisoning and procedural complications) | 2/9333 | 0/9291
Overdose (Injury, poisoning and procedural complications) | 2/9333 | 0/9291
Postoperative Thrombosis (Injury, poisoning and procedural complications) | 1/9333 | 2/9291
Procedural Hypotension (Injury, poisoning and procedural complications) | 0/9333 | 2/9291
Renal Injury (Injury, poisoning and procedural complications) | 1/9333 | 2/9291
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 2/9333 | 2/9291
Stent Occlusion (Injury, poisoning and procedural complications) | 1/9333 | 2/9291
Traumatic Haemorrhage (Injury, poisoning and procedural complications) | 1/9333 | 2/9291
Upper Limb Fracture (Injury, poisoning and procedural complications) | 1/9333 | 2/9291
Vascular Graft Occlusion (Injury, poisoning and procedural complications) | 2/9333 | 0/9291
Anaemia Postoperative (Injury, poisoning and procedural complications) | 0/9333 | 1/9291
Ankle Fracture (Injury, poisoning and procedural complications) | 1/9333 | 0/9291
Brain Contusion (Injury, poisoning and procedural complications) | 1/9333 | 0/9291
Cardiac Pacemaker Malfunction (Injury, poisoning and procedural complications) | 1/9333 | 0/9291
Cardiac Procedure Complication (Injury, poisoning and procedural complications) | 1/9333 | 0/9291
Chest Injury (Injury, poisoning and procedural complications) | 1/9333 | 0/9291
Contrast Media Reaction (Injury, poisoning and procedural complications) | 0/9333 | 1/9291
Contusion (Injury, poisoning and procedural complications) | 0/9333 | 1/9291
Coronary Artery Reocclusion (Injury, poisoning and procedural complications) | 0/9333 | 1/9291
Device Breakage (Injury, poisoning and procedural complications) | 1/9333 | 1/9291
Device Dislocation (Injury, poisoning and procedural complications) | 1/9333 | 0/9291
Device Malfunction (Injury, poisoning and procedural complications) | 1/9333 | 1/9291
Device Migration (Injury, poisoning and procedural complications) | 0/9333 | 1/9291
Fat Embolism (Injury, poisoning and procedural complications) | 1/9333 | 0/9291
Forearm Fracture (Injury, poisoning and procedural complications) | 1/9333 | 0/9291
Fracture (Injury, poisoning and procedural complications) | 1/9333 | 0/9291
Fractured Ischium (Injury, poisoning and procedural complications) | 0/9333 | 1/9291
Implantable Defibrillator Malfunction (Injury, poisoning and procedural complications) | 0/9333 | 1/9291
Incision Site Haemorrhage (Injury, poisoning and procedural complications) | 0/9333 | 1/9291
Incisional Hernia (Injury, poisoning and procedural complications) | 0/9333 | 1/9291
Joint Dislocation (Injury, poisoning and procedural complications) | 1/9333 | 1/9291
Joint Injury (Injury, poisoning and procedural complications) | 0/9333 | 1/9291
Joint Sprain (Injury, poisoning and procedural complications) | 0/9333 | 1/9291
Lumbar Vertebral Fracture (Injury, poisoning and procedural complications) | 0/9333 | 1/9291
Meniscus Lesion (Injury, poisoning and procedural complications) | 1/9333 | 0/9291
Open Wound (Injury, poisoning and procedural complications) | 1/9333 | 0/9291
Pelvic Fracture (Injury, poisoning and procedural complications) | 1/9333 | 1/9291
Post Procedural Haematuria (Injury, poisoning and procedural complications) | 1/9333 | 0/9291
Procedural Complication (Injury, poisoning and procedural complications) | 0/9333 | 1/9291
Radius Fracture (Injury, poisoning and procedural complications) | 1/9333 | 1/9291
Rib Fracture (Injury, poisoning and procedural complications) | 0/9333 | 1/9291
Road Traffic Accident (Injury, poisoning and procedural complications) | 1/9333 | 0/9291
Scrotal Haematoma (Injury, poisoning and procedural complications) | 1/9333 | 0/9291
Suture Rupture (Injury, poisoning and procedural complications) | 0/9333 | 1/9291
Tendon Rupture (Injury, poisoning and procedural complications) | 0/9333 | 1/9291
Thermal Burn (Injury, poisoning and procedural complications) | 1/9333 | 0/9291
Tibia Fracture (Injury, poisoning and procedural complications) | 1/9333 | 0/9291
Tracheal Haemorrhage (Injury, poisoning and procedural complications) | 0/9333 | 1/9291
Tracheal Obstruction (Injury, poisoning and procedural complications) | 0/9333 | 1/9291
Transfusion Reaction (Injury, poisoning and procedural complications) | 0/9333 | 1/9291
Traumatic Intracranial Haemorrhage (Injury, poisoning and procedural complications) | 1/9333 | 0/9291
Ulna Fracture (Injury, poisoning and procedural complications) | 0/9333 | 1/9291
Urinary Bladder Rupture (Injury, poisoning and procedural complications) | 0/9333 | 1/9291
Urinary Retention Postoperative (Injury, poisoning and procedural complications) | 1/9333 | 0/9291
Vascular Procedure Complication (Injury, poisoning and procedural complications) | 1/9333 | 0/9291
Vascular Pseudoaneurysm Ruptured (Injury, poisoning and procedural complications) | 1/9333 | 0/9291
Vertebral Injury (Injury, poisoning and procedural complications) | 1/9333 | 0/9291
Weaning Failure (Injury, poisoning and procedural complications) | 1/9333 | 0/9291
Wound Complication (Injury, poisoning and procedural complications) | 0/9333 | 1/9291
Haemoglobin Decreased (Injury, poisoning and procedural complications) | 6/9333 | 8/9291
Aspartate Aminotransferase Increased (Injury, poisoning and procedural complications) | 1/9333 | 4/9291
Alanine Aminotransferase Increased (Injury, poisoning and procedural complications) | 1/9333 | 3/9291
Blood Pressure Increased (Injury, poisoning and procedural complications) | 3/9333 | 3/9291
Liver Function Test Abnormal (Injury, poisoning and procedural complications) | 2/9333 | 3/9291
Angiogram (Injury, poisoning and procedural complications) | 2/9333 | 0/9291
Blood Glucose Increased (Injury, poisoning and procedural complications) | 2/9333 | 1/9291
Blood Potassium Increased (Injury, poisoning and procedural complications) | 0/9333 | 2/9291
Body Temperature Increased (Injury, poisoning and procedural complications) | 2/9333 | 0/9291
Hepatic Enzyme Increased (Injury, poisoning and procedural complications) | 2/9333 | 2/9291
International Normalised Ratio Increased (Injury, poisoning and procedural complications) | 1/9333 | 2/9291
Troponin Increased (Injury, poisoning and procedural complications) | 1/9333 | 2/9291
Antiphospholipid Antibodies (Injury, poisoning and procedural complications) | 0/9333 | 1/9291
Blood Creatine Phosphokinase Increased (Injury, poisoning and procedural complications) | 1/9333 | 1/9291
Blood Creatinine Increased (Injury, poisoning and procedural complications) | 1/9333 | 0/9291
Blood Potassium Decreased (Injury, poisoning and procedural complications) | 1/9333 | 0/9291
Blood Pressure Decreased (Injury, poisoning and procedural complications) | 1/9333 | 0/9291
Blood Sodium Decreased (Injury, poisoning and procedural complications) | 1/9333 | 0/9291
Blood Urine Present (Injury, poisoning and procedural complications) | 1/9333 | 0/9291
C-Reactive Protein Increased (Injury, poisoning and procedural complications) | 1/9333 | 0/9291
Cardiac Enzymes Increased (Injury, poisoning and procedural complications) | 1/9333 | 0/9291
Cardiac Stress Test Abnormal (Injury, poisoning and procedural complications) | 1/9333 | 0/9291
Electrocardiogram Qt Prolonged (Injury, poisoning and procedural complications) | 1/9333 | 1/9291
Electrocardiogram T Wave Inversion (Injury, poisoning and procedural complications) | 1/9333 | 0/9291
Fibrin D Dimer Increased (Injury, poisoning and procedural complications) | 0/9333 | 1/9291
Heart Rate Increased (Injury, poisoning and procedural complications) | 0/9333 | 1/9291
Intraocular Pressure Increased (Injury, poisoning and procedural complications) | 0/9333 | 1/9291
Occult Blood (Injury, poisoning and procedural complications) | 1/9333 | 0/9291
Pancreatic Enzymes Increased (Injury, poisoning and procedural complications) | 0/9333 | 1/9291
Platelet Count Decreased (Injury, poisoning and procedural complications) | 0/9333 | 1/9291
Prostatic Specific Antigen Abnormal (Injury, poisoning and procedural complications) | 1/9333 | 0/9291
Prostatic Specific Antigen Increased (Injury, poisoning and procedural complications) | 1/9333 | 0/9291
Weight Decreased (Injury, poisoning and procedural complications) | 1/9333 | 1/9291
Dehydration (Metabolism and nutrition disorders) | 11/9333 | 5/9291
Hypoglycaemia (Metabolism and nutrition disorders) | 11/9333 | 8/9291
Diabetes Mellitus Inadequate Control (Metabolism and nutrition disorders) | 3/9333 | 9/9291
Diabetes Mellitus (Metabolism and nutrition disorders) | 6/9333 | 7/9291
Hyperglycaemia (Metabolism and nutrition disorders) | 7/9333 | 2/9291
Hyperkalaemia (Metabolism and nutrition disorders) | 1/9333 | 4/9291
Anorexia (Metabolism and nutrition disorders) | 3/9333 | 0/9291
Hyponatraemia (Metabolism and nutrition disorders) | 3/9333 | 1/9291
Diabetic Ketoacidosis (Metabolism and nutrition disorders) | 2/9333 | 1/9291
Fluid Overload (Metabolism and nutrition disorders) | 0/9333 | 2/9291
Gout (Metabolism and nutrition disorders) | 2/9333 | 2/9291
Metabolic Acidosis (Metabolism and nutrition disorders) | 0/9333 | 2/9291
Metabolic Disorder (Metabolism and nutrition disorders) | 0/9333 | 2/9291
Type 2 Diabetes Mellitus (Metabolism and nutrition disorders) | 2/9333 | 2/9291
Diabetic Foot (Metabolism and nutrition disorders) | 1/9333 | 0/9291
Electrolyte Depletion (Metabolism and nutrition disorders) | 0/9333 | 1/9291
Failure To Thrive (Metabolism and nutrition disorders) | 0/9333 | 1/9291
Hyperosmolar State (Metabolism and nutrition disorders) | 0/9333 | 1/9291
Hypokalaemia (Metabolism and nutrition disorders) | 1/9333 | 1/9291
Hypovolaemia (Metabolism and nutrition disorders) | 1/9333 | 0/9291
Ketoacidosis (Metabolism and nutrition disorders) | 1/9333 | 0/9291
Metabolic Syndrome (Metabolism and nutrition disorders) | 0/9333 | 1/9291
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 15/9333 | 16/9291
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 7/9333 | 5/9291
Back Pain (Musculoskeletal and connective tissue disorders) | 3/9333 | 6/9291
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 5/9333 | 4/9291
Arthralgia (Musculoskeletal and connective tissue disorders) | 3/9333 | 4/9291
Myalgia (Musculoskeletal and connective tissue disorders) | 3/9333 | 3/9291
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 3/9333 | 2/9291
Arthritis (Musculoskeletal and connective tissue disorders) | 2/9333 | 2/9291
Bone Pain (Musculoskeletal and connective tissue disorders) | 1/9333 | 2/9291
Bursitis (Musculoskeletal and connective tissue disorders) | 2/9333 | 1/9291
Costochondritis (Musculoskeletal and connective tissue disorders) | 2/9333 | 1/9291
Gouty Arthritis (Musculoskeletal and connective tissue disorders) | 2/9333 | 0/9291
Myalgia Intercostal (Musculoskeletal and connective tissue disorders) | 2/9333 | 0/9291
Neck Pain (Musculoskeletal and connective tissue disorders) | 1/9333 | 2/9291
Chondropathy (Musculoskeletal and connective tissue disorders) | 0/9333 | 1/9291
Dupuytren's Contracture (Musculoskeletal and connective tissue disorders) | 0/9333 | 1/9291
Groin Pain (Musculoskeletal and connective tissue disorders) | 1/9333 | 0/9291
Intervertebral Disc Degeneration (Musculoskeletal and connective tissue disorders) | 0/9333 | 1/9291
Intervertebral Disc Disorder (Musculoskeletal and connective tissue disorders) | 0/9333 | 1/9291
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 1/9333 | 1/9291
Joint Swelling (Musculoskeletal and connective tissue disorders) | 1/9333 | 0/9291
Lumbar Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 0/9333 | 1/9291
Monarthritis (Musculoskeletal and connective tissue disorders) | 1/9333 | 0/9291
Muscle Tightness (Musculoskeletal and connective tissue disorders) | 1/9333 | 0/9291
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1/9333 | 1/9291
Myositis (Musculoskeletal and connective tissue disorders) | 0/9333 | 1/9291
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 1/9333 | 0/9291
Osteolysis (Musculoskeletal and connective tissue disorders) | 1/9333 | 0/9291
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0/9333 | 1/9291
Pain In Jaw (Musculoskeletal and connective tissue disorders) | 1/9333 | 0/9291
Pathological Fracture (Musculoskeletal and connective tissue disorders) | 0/9333 | 1/9291
Polyarthritis (Musculoskeletal and connective tissue disorders) | 1/9333 | 0/9291
Polymyalgia Rheumatica (Musculoskeletal and connective tissue disorders) | 1/9333 | 0/9291
Polymyositis (Musculoskeletal and connective tissue disorders) | 0/9333 | 1/9291
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1/9333 | 1/9291
Rheumatoid Arthritis (Musculoskeletal and connective tissue disorders) | 1/9333 | 0/9291
Spinal Disorder (Musculoskeletal and connective tissue disorders) | 1/9333 | 0/9291
Spinal Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0/9333 | 1/9291
Wrist Deformity (Musculoskeletal and connective tissue disorders) | 0/9333 | 1/9291
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 10/9333 | 3/9291
Lung Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6/9333 | 10/9291
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3/9333 | 9/9291
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6/9333 | 8/9291
Lung Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7/9333 | 5/9291
Bladder Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2/9333 | 6/9291
Colon Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/9333 | 5/9291
Renal Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5/9333 | 3/9291
Bladder Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/9333 | 3/9291
Brain Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/9333 | 3/9291
Bronchial Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/9333 | 3/9291
Gastric Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3/9333 | 3/9291
Metastases To Liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/9333 | 3/9291
Rectal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3/9333 | 2/9291
Bladder Transitional Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2/9333 | 1/9291
Chronic Lymphocytic Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2/9333 | 1/9291
Gastrointestinal Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2/9333 | 0/9291
Hepatic Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2/9333 | 1/9291
Laryngeal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/9333 | 2/9291
Lung Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2/9333 | 0/9291
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2/9333 | 1/9291
Malignant Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/9333 | 2/9291
Metastases To Bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/9333 | 2/9291
Metastases To Lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/9333 | 2/9291
Metastatic Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2/9333 | 0/9291
Oesophageal Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/9333 | 2/9291
Ovarian Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2/9333 | 1/9291
Renal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2/9333 | 1/9291
Abdominal Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/9333 | 0/9291
Acute Myeloid Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/9333 | 0/9291
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/9333 | 0/9291
Adenocarcinoma Pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/9333 | 1/9291
B-Cell Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/9333 | 1/9291
Benign Duodenal Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/9333 | 0/9291
Benign Neoplasm Of Skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/9333 | 1/9291
Benign Uterine Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/9333 | 1/9291
Bladder Cancer Recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/9333 | 1/9291
Bone Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/9333 | 1/9291
Brain Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/9333 | 1/9291
Breast Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/9333 | 0/9291
Bronchial Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/9333 | 0/9291
Carcinoid Tumour Of The Caecum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/9333 | 1/9291
Carcinoid Tumour Of The Duodenum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/9333 | 1/9291
Chronic Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/9333 | 1/9291
Colon Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/9333 | 1/9291
Colorectal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/9333 | 1/9291
Endometrial Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/9333 | 0/9291
Extranodal Marginal Zone B-Cell Lymphoma (Malt Type) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/9333 | 0/9291
Gastric Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/9333 | 0/9291
Gastrointestinal Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/9333 | 1/9291
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/9333 | 0/9291
Haemangioma Of Liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/9333 | 0/9291
Hepatic Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/9333 | 1/9291
Intestinal Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/9333 | 1/9291
Lip And/Or Oral Cavity Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/9333 | 1/9291
Lung Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/9333 | 0/9291
Lymphangiosis Carcinomatosa (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/9333 | 1/9291
Lymphocytic Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/9333 | 0/9291
Malignant Pleural Effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/9333 | 0/9291
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/9333 | 0/9291
Metastases To Central Nervous System (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/9333 | 1/9291
Metastases To Lymph Nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/9333 | 0/9291
Myelodysplastic Syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/9333 | 1/9291
Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/9333 | 1/9291
Neoplasm Prostate (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/9333 | 1/9291
Nipple Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/9333 | 1/9291
Pancreatic Carcinoma Recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/9333 | 0/9291
Pleural Mesothelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/9333 | 1/9291
Polycythaemia Vera (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/9333 | 0/9291
Prostate Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/9333 | 1/9291
Prostate Cancer Recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/9333 | 0/9291
Prostatic Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/9333 | 1/9291
Rectal Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/9333 | 0/9291
Renal Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/9333 | 1/9291
Retroperitoneal Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/9333 | 1/9291
Small Cell Lung Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/9333 | 1/9291
Small Cell Lung Cancer Stage Unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/9333 | 1/9291
Spinal Cord Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/9333 | 1/9291
Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/9333 | 1/9291
Testis Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/9333 | 0/9291
Thyroid Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/9333 | 0/9291
Thyroid Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/9333 | 0/9291
Thyroid Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/9333 | 1/9291
Tongue Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/9333 | 1/9291
Transitional Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/9333 | 1/9291
Uterine Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/9333 | 0/9291
Cerebrovascular Accident (Nervous system disorders) | 75/9333 | 50/9291
Syncope (Nervous system disorders) | 32/9333 | 30/9291
Ischaemic Stroke (Nervous system disorders) | 20/9333 | 28/9291
Transient Ischaemic Attack (Nervous system disorders) | 19/9333 | 23/9291
Dizziness (Nervous system disorders) | 13/9333 | 7/9291
Cerebral Haemorrhage (Nervous system disorders) | 9/9333 | 3/9291
Cerebral Infarction (Nervous system disorders) | 7/9333 | 8/9291
Presyncope (Nervous system disorders) | 8/9333 | 2/9291
Haemorrhagic Stroke (Nervous system disorders) | 6/9333 | 7/9291
Headache (Nervous system disorders) | 6/9333 | 3/9291
Haemorrhage Intracranial (Nervous system disorders) | 5/9333 | 2/9291
Paraesthesia (Nervous system disorders) | 5/9333 | 4/9291
Hemiparesis (Nervous system disorders) | 4/9333 | 2/9291
Loss Of Consciousness (Nervous system disorders) | 4/9333 | 2/9291
Parkinson's Disease (Nervous system disorders) | 1/9333 | 4/9291
Subarachnoid Haemorrhage (Nervous system disorders) | 4/9333 | 2/9291
Syncope Vasovagal (Nervous system disorders) | 4/9333 | 2/9291
Carotid Artery Stenosis (Nervous system disorders) | 3/9333 | 2/9291
Convulsion (Nervous system disorders) | 3/9333 | 3/9291
Depressed Level Of Consciousness (Nervous system disorders) | 0/9333 | 3/9291
Hypoaesthesia (Nervous system disorders) | 2/9333 | 3/9291
Hypotonia (Nervous system disorders) | 3/9333 | 0/9291
Migraine (Nervous system disorders) | 3/9333 | 1/9291
Altered State Of Consciousness (Nervous system disorders) | 0/9333 | 2/9291
Brain Stem Ischaemia (Nervous system disorders) | 0/9333 | 2/9291
Cerebral Ischaemia (Nervous system disorders) | 2/9333 | 1/9291
Cerebrovascular Disorder (Nervous system disorders) | 0/9333 | 2/9291
Dementia (Nervous system disorders) | 0/9333 | 2/9291
Encephalopathy (Nervous system disorders) | 2/9333 | 1/9291
Hypoxic Encephalopathy (Nervous system disorders) | 0/9333 | 2/9291
Neuralgia (Nervous system disorders) | 2/9333 | 0/9291
Partial Seizures (Nervous system disorders) | 2/9333 | 0/9291
Balance Disorder (Nervous system disorders) | 1/9333 | 0/9291
Brain Oedema (Nervous system disorders) | 1/9333 | 0/9291
Brain Stem Infarction (Nervous system disorders) | 0/9333 | 1/9291
Brain Stem Stroke (Nervous system disorders) | 0/9333 | 1/9291
Carotid Artery Disease (Nervous system disorders) | 0/9333 | 1/9291
Carotid Artery Occlusion (Nervous system disorders) | 0/9333 | 1/9291
Carotid Artery Thrombosis (Nervous system disorders) | 0/9333 | 1/9291
Carotid Sinus Syndrome (Nervous system disorders) | 1/9333 | 0/9291
Central Nervous System Lesion (Nervous system disorders) | 1/9333 | 0/9291
Cerebellar Infarction (Nervous system disorders) | 1/9333 | 0/9291
Cerebral Atrophy (Nervous system disorders) | 0/9333 | 1/9291
Cerebral Disorder (Nervous system disorders) | 1/9333 | 0/9291
Cerebrovascular Insufficiency (Nervous system disorders) | 1/9333 | 0/9291
Cervicobrachial Syndrome (Nervous system disorders) | 0/9333 | 1/9291
Cognitive Disorder (Nervous system disorders) | 0/9333 | 1/9291
Complex Partial Seizures (Nervous system disorders) | 0/9333 | 1/9291
Diabetic Hyperosmolar Coma (Nervous system disorders) | 1/9333 | 0/9291
Diabetic Neuropathy (Nervous system disorders) | 1/9333 | 0/9291
Dysphasia (Nervous system disorders) | 0/9333 | 1/9291
Embolic Cerebral Infarction (Nervous system disorders) | 1/9333 | 0/9291
Encephalitis (Nervous system disorders) | 0/9333 | 1/9291
Epilepsy (Nervous system disorders) | 1/9333 | 1/9291
Extrapyramidal Disorder (Nervous system disorders) | 0/9333 | 1/9291
Facial Paresis (Nervous system disorders) | 1/9333 | 0/9291
Febrile Convulsion (Nervous system disorders) | 1/9333 | 0/9291
Haemorrhagic Cerebral Infarction (Nervous system disorders) | 1/9333 | 0/9291
Hepatic Encephalopathy (Nervous system disorders) | 0/9333 | 1/9291
Intracranial Haematoma (Nervous system disorders) | 0/9333 | 1/9291
Ischaemic Cerebral Infarction (Nervous system disorders) | 1/9333 | 1/9291
Lacunar Infarction (Nervous system disorders) | 1/9333 | 0/9291
Lumbar Radiculopathy (Nervous system disorders) | 1/9333 | 0/9291
Mental Impairment (Nervous system disorders) | 0/9333 | 1/9291
Myelitis Transverse (Nervous system disorders) | 0/9333 | 1/9291
Narcolepsy (Nervous system disorders) | 0/9333 | 1/9291
Parkinsonism (Nervous system disorders) | 0/9333 | 1/9291
Phrenic Nerve Paralysis (Nervous system disorders) | 1/9333 | 0/9291
Post Herpetic Neuralgia (Nervous system disorders) | 0/9333 | 1/9291
Progressive Supranuclear Palsy (Nervous system disorders) | 0/9333 | 1/9291
Psychomotor Hyperactivity (Nervous system disorders) | 0/9333 | 1/9291
Sciatica (Nervous system disorders) | 0/9333 | 1/9291
Speech Disorder (Nervous system disorders) | 1/9333 | 0/9291
Spinal Cord Compression (Nervous system disorders) | 0/9333 | 1/9291
Spinal Cord Disorder (Nervous system disorders) | 1/9333 | 0/9291
Thalamus Haemorrhage (Nervous system disorders) | 1/9333 | 0/9291
Thrombotic Stroke (Nervous system disorders) | 1/9333 | 0/9291
Vascular Encephalopathy (Nervous system disorders) | 1/9333 | 0/9291
Vertebrobasilar Insufficiency (Nervous system disorders) | 1/9333 | 1/9291
Vith Nerve Paralysis (Nervous system disorders) | 0/9333 | 1/9291
Vocal Cord Paresis (Nervous system disorders) | 1/9333 | 0/9291
Anxiety (Psychiatric disorders) | 9/9333 | 6/9291
Depression (Psychiatric disorders) | 9/9333 | 7/9291
Confusional State (Psychiatric disorders) | 4/9333 | 2/9291
Suicide Attempt (Psychiatric disorders) | 1/9333 | 2/9291
Acute Stress Disorder (Psychiatric disorders) | 1/9333 | 1/9291
Agitation (Psychiatric disorders) | 1/9333 | 0/9291
Alcohol Abuse (Psychiatric disorders) | 1/9333 | 0/9291
Alcoholism (Psychiatric disorders) | 0/9333 | 1/9291
Anxiety Disorder (Psychiatric disorders) | 1/9333 | 1/9291
Completed Suicide (Psychiatric disorders) | 1/9333 | 1/9291
Delirium (Psychiatric disorders) | 1/9333 | 1/9291
Drug Abuse (Psychiatric disorders) | 0/9333 | 1/9291
Insomnia (Psychiatric disorders) | 1/9333 | 0/9291
Mania (Psychiatric disorders) | 1/9333 | 0/9291
Mental Disorder (Psychiatric disorders) | 0/9333 | 1/9291
Nervousness (Psychiatric disorders) | 0/9333 | 1/9291
Neurosis (Psychiatric disorders) | 0/9333 | 1/9291
Panic Attack (Psychiatric disorders) | 1/9333 | 0/9291
Post-Traumatic Amnestic Disorder (Psychiatric disorders) | 1/9333 | 0/9291
Psychotic Disorder (Psychiatric disorders) | 1/9333 | 0/9291
Schizophrenia, Paranoid Type (Psychiatric disorders) | 0/9333 | 1/9291
Sleep Disorder (Psychiatric disorders) | 1/9333 | 0/9291
Suicidal Ideation (Psychiatric disorders) | 1/9333 | 1/9291
Tension (Psychiatric disorders) | 1/9333 | 0/9291
Transient Psychosis (Psychiatric disorders) | 1/9333 | 0/9291
Renal Failure Acute (Renal and urinary disorders) | 34/9333 | 25/9291
Renal Failure (Renal and urinary disorders) | 25/9333 | 24/9291
Haematuria (Renal and urinary disorders) | 15/9333 | 10/9291
Renal Failure Chronic (Renal and urinary disorders) | 7/9333 | 7/9291
Urinary Retention (Renal and urinary disorders) | 3/9333 | 7/9291
Renal Impairment (Renal and urinary disorders) | 5/9333 | 4/9291
Calculus Ureteric (Renal and urinary disorders) | 2/9333 | 4/9291
Calculus Urinary (Renal and urinary disorders) | 0/9333 | 3/9291
Haemorrhage Urinary Tract (Renal and urinary disorders) | 3/9333 | 1/9291
Nephrolithiasis (Renal and urinary disorders) | 3/9333 | 3/9291
Nephropathy Toxic (Renal and urinary disorders) | 3/9333 | 2/9291
Renal Artery Stenosis (Renal and urinary disorders) | 2/9333 | 3/9291
Renal Colic (Renal and urinary disorders) | 3/9333 | 1/9291
Azotaemia (Renal and urinary disorders) | 2/9333 | 1/9291
Urinary Bladder Haemorrhage (Renal and urinary disorders) | 2/9333 | 0/9291
Urinary Bladder Polyp (Renal and urinary disorders) | 0/9333 | 2/9291
Anuria (Renal and urinary disorders) | 1/9333 | 1/9291
Bladder Mass (Renal and urinary disorders) | 1/9333 | 0/9291
Bladder Prolapse (Renal and urinary disorders) | 0/9333 | 1/9291
Bladder Tamponade (Renal and urinary disorders) | 1/9333 | 1/9291
Calculus Bladder (Renal and urinary disorders) | 0/9333 | 1/9291
Calculus Urethral (Renal and urinary disorders) | 0/9333 | 1/9291
Cystitis Haemorrhagic (Renal and urinary disorders) | 0/9333 | 1/9291
Cystitis Noninfective (Renal and urinary disorders) | 0/9333 | 1/9291
Dysuria (Renal and urinary disorders) | 1/9333 | 0/9291
Glomerulonephritis (Renal and urinary disorders) | 1/9333 | 0/9291
Glomerulonephritis Membranous (Renal and urinary disorders) | 0/9333 | 1/9291
Glomerulonephritis Minimal Lesion (Renal and urinary disorders) | 0/9333 | 1/9291
Hydronephrosis (Renal and urinary disorders) | 0/9333 | 1/9291
Nephritis Autoimmune (Renal and urinary disorders) | 1/9333 | 0/9291
Nephrotic Syndrome (Renal and urinary disorders) | 0/9333 | 1/9291
Obstructive Uropathy (Renal and urinary disorders) | 0/9333 | 1/9291
Oliguria (Renal and urinary disorders) | 1/9333 | 0/9291
Renal Artery Thrombosis (Renal and urinary disorders) | 1/9333 | 0/9291
Renal Disorder (Renal and urinary disorders) | 1/9333 | 0/9291
Renal Haemorrhage (Renal and urinary disorders) | 1/9333 | 0/9291
Renal Mass (Renal and urinary disorders) | 1/9333 | 1/9291
Urethral Haemorrhage (Renal and urinary disorders) | 1/9333 | 0/9291
Urinary Incontinence (Renal and urinary disorders) | 0/9333 | 1/9291
Urinary Tract Obstruction (Renal and urinary disorders) | 0/9333 | 1/9291
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 5/9333 | 3/9291
Epididymitis (Reproductive system and breast disorders) | 3/9333 | 1/9291
Prostatitis (Reproductive system and breast disorders) | 1/9333 | 2/9291
Balanitis (Reproductive system and breast disorders) | 0/9333 | 1/9291
Cervical Dysplasia (Reproductive system and breast disorders) | 1/9333 | 0/9291
Menometrorrhagia (Reproductive system and breast disorders) | 0/9333 | 1/9291
Ovarian Cyst (Reproductive system and breast disorders) | 0/9333 | 1/9291
Prostatic Haemorrhage (Reproductive system and breast disorders) | 1/9333 | 1/9291
Prostatism (Reproductive system and breast disorders) | 1/9333 | 0/9291
Spermatocele (Reproductive system and breast disorders) | 0/9333 | 1/9291
Uterine Haemorrhage (Reproductive system and breast disorders) | 1/9333 | 0/9291
Vaginal Haemorrhage (Reproductive system and breast disorders) | 0/9333 | 1/9291
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 75/9333 | 50/9291
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 33/9333 | 53/9291
Acute Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 20/9333 | 32/9291
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 31/9333 | 20/9291
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 22/9333 | 17/9291
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 21/9333 | 19/9291
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 16/9333 | 16/9291
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 15/9333 | 9/9291
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3/9333 | 9/9291
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 7/9333 | 8/9291
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 5/9333 | 6/9291
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 3/9333 | 6/9291
Asthma (Respiratory, thoracic and mediastinal disorders) | 5/9333 | 3/9291
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 2/9333 | 5/9291
Pulmonary Congestion (Respiratory, thoracic and mediastinal disorders) | 5/9333 | 3/9291
Acute Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 4/9333 | 3/9291
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0/9333 | 3/9291
Cough (Respiratory, thoracic and mediastinal disorders) | 3/9333 | 0/9291
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 3/9333 | 2/9291
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0/9333 | 3/9291
Pleuritic Pain (Respiratory, thoracic and mediastinal disorders) | 0/9333 | 3/9291
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3/9333 | 0/9291
Pulmonary Mass (Respiratory, thoracic and mediastinal disorders) | 3/9333 | 0/9291
Respiratory Arrest (Respiratory, thoracic and mediastinal disorders) | 2/9333 | 3/9291
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 2/9333 | 1/9291
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 2/9333 | 1/9291
Lung Disorder (Respiratory, thoracic and mediastinal disorders) | 2/9333 | 1/9291
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 2/9333 | 2/9291
Pulmonary Haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1/9333 | 2/9291
Alveolitis Fibrosing (Respiratory, thoracic and mediastinal disorders) | 0/9333 | 1/9291
Apnoea (Respiratory, thoracic and mediastinal disorders) | 0/9333 | 1/9291
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1/9333 | 0/9291
Brain Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0/9333 | 1/9291
Bronchial Haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1/9333 | 0/9291
Bronchial Obstruction (Respiratory, thoracic and mediastinal disorders) | 1/9333 | 0/9291
Bronchitis Chronic (Respiratory, thoracic and mediastinal disorders) | 1/9333 | 0/9291
Dyspnoea Paroxysmal Nocturnal (Respiratory, thoracic and mediastinal disorders) | 0/9333 | 1/9291
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1/9333 | 0/9291
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0/9333 | 1/9291
Interstitial Lung Disease (Respiratory, thoracic and mediastinal disorders) | 0/9333 | 1/9291
Laryngeal Leukoplakia (Respiratory, thoracic and mediastinal disorders) | 1/9333 | 0/9291
Laryngeal Oedema (Respiratory, thoracic and mediastinal disorders) | 1/9333 | 1/9291
Laryngeal Stenosis (Respiratory, thoracic and mediastinal disorders) | 0/9333 | 1/9291
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 1/9333 | 0/9291
Lower Respiratory Tract Inflammation (Respiratory, thoracic and mediastinal disorders) | 1/9333 | 0/9291
Lung Consolidation (Respiratory, thoracic and mediastinal disorders) | 1/9333 | 0/9291
Mediastinal Haematoma (Respiratory, thoracic and mediastinal disorders) | 0/9333 | 1/9291
Mediastinal Haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0/9333 | 1/9291
Nasal Polyps (Respiratory, thoracic and mediastinal disorders) | 0/9333 | 1/9291
Nocturnal Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1/9333 | 0/9291
Pulmonary Alveolar Haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1/9333 | 0/9291
Pulmonary Fibrosis (Respiratory, thoracic and mediastinal disorders) | 1/9333 | 0/9291
Pulmonary Haematoma (Respiratory, thoracic and mediastinal disorders) | 0/9333 | 1/9291
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 1/9333 | 0/9291
Respiratory Tract Haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1/9333 | 1/9291
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1/9333 | 0/9291
Systemic Sclerosis Pulmonary (Respiratory, thoracic and mediastinal disorders) | 0/9333 | 1/9291
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1/9333 | 0/9291
Thoracic Haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0/9333 | 1/9291
Tonsillar Disorder (Respiratory, thoracic and mediastinal disorders) | 1/9333 | 0/9291
Tracheal Stenosis (Respiratory, thoracic and mediastinal disorders) | 0/9333 | 1/9291
Vocal Cord Polyp (Respiratory, thoracic and mediastinal disorders) | 1/9333 | 1/9291
Wegener's Granulomatosis (Respiratory, thoracic and mediastinal disorders) | 0/9333 | 1/9291
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1/9333 | 0/9291
Dermatitis Allergic (Skin and subcutaneous tissue disorders) | 1/9333 | 6/9291
Angioedema (Skin and subcutaneous tissue disorders) | 3/9333 | 4/9291
Rash (Skin and subcutaneous tissue disorders) | 4/9333 | 3/9291
Urticaria (Skin and subcutaneous tissue disorders) | 3/9333 | 4/9291
Pruritus (Skin and subcutaneous tissue disorders) | 1/9333 | 3/9291
Skin Ulcer (Skin and subcutaneous tissue disorders) | 3/9333 | 0/9291
Decubitus Ulcer (Skin and subcutaneous tissue disorders) | 2/9333 | 0/9291
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2/9333 | 0/9291
Skin Necrosis (Skin and subcutaneous tissue disorders) | 2/9333 | 1/9291
Alopecia (Skin and subcutaneous tissue disorders) | 0/9333 | 1/9291
Blister (Skin and subcutaneous tissue disorders) | 0/9333 | 1/9291
Dermatitis (Skin and subcutaneous tissue disorders) | 1/9333 | 0/9291
Dermatomyositis (Skin and subcutaneous tissue disorders) | 1/9333 | 0/9291
Dry Gangrene (Skin and subcutaneous tissue disorders) | 1/9333 | 1/9291
Eczema Nummular (Skin and subcutaneous tissue disorders) | 0/9333 | 1/9291
Erythema (Skin and subcutaneous tissue disorders) | 0/9333 | 1/9291
Hypoaesthesia Facial (Skin and subcutaneous tissue disorders) | 0/9333 | 1/9291
Increased Tendency To Bruise (Skin and subcutaneous tissue disorders) | 1/9333 | 0/9291
Leukocytoclastic Vasculitis (Skin and subcutaneous tissue disorders) | 0/9333 | 1/9291
Pruritus Generalised (Skin and subcutaneous tissue disorders) | 1/9333 | 0/9291
Rash Erythematous (Skin and subcutaneous tissue disorders) | 1/9333 | 0/9291
Rash Generalised (Skin and subcutaneous tissue disorders) | 1/9333 | 0/9291
Seborrhoeic Dermatitis (Skin and subcutaneous tissue disorders) | 0/9333 | 1/9291
Skin Inflammation (Skin and subcutaneous tissue disorders) | 1/9333 | 0/9291
Cardiac Pacemaker Insertion (Surgical and medical procedures) | 1/9333 | 0/9291
Coronary Artery Bypass (Surgical and medical procedures) | 1/9333 | 1/9291
Implantable Defibrillator Insertion (Surgical and medical procedures) | 0/9333 | 1/9291
Leg Amputation (Surgical and medical procedures) | 1/9333 | 0/9291
Thoracic Cavity Drainage (Surgical and medical procedures) | 0/9333 | 1/9291
Hypertension (Vascular disorders) | 17/9333 | 24/9291
Hypotension (Vascular disorders) | 18/9333 | 21/9291
Hypertensive Crisis (Vascular disorders) | 7/9333 | 12/9291
Peripheral Ischaemia (Vascular disorders) | 10/9333 | 7/9291
Haematoma (Vascular disorders) | 3/9333 | 8/9291
Aortic Aneurysm (Vascular disorders) | 0/9333 | 7/9291
Shock (Vascular disorders) | 7/9333 | 3/9291
Deep Vein Thrombosis (Vascular disorders) | 6/9333 | 6/9291
Intermittent Claudication (Vascular disorders) | 6/9333 | 6/9291
Accelerated Hypertension (Vascular disorders) | 1/9333 | 5/9291
Arterial Thrombosis Limb (Vascular disorders) | 5/9333 | 4/9291
Peripheral Arterial Occlusive Disease (Vascular disorders) | 4/9333 | 5/9291
Peripheral Vascular Disorder (Vascular disorders) | 5/9333 | 3/9291
Aortic Dissection (Vascular disorders) | 2/9333 | 4/9291
Arterial Thrombosis (Vascular disorders) | 1/9333 | 4/9291
Circulatory Collapse (Vascular disorders) | 4/9333 | 0/9291
Orthostatic Hypotension (Vascular disorders) | 4/9333 | 3/9291
Aortic Stenosis (Vascular disorders) | 0/9333 | 3/9291
Arteriosclerosis (Vascular disorders) | 3/9333 | 3/9291
Femoral Artery Aneurysm (Vascular disorders) | 1/9333 | 3/9291
Haemorrhage (Vascular disorders) | 2/9333 | 3/9291
Hypertensive Emergency (Vascular disorders) | 3/9333 | 3/9291
Hypovolaemic Shock (Vascular disorders) | 3/9333 | 2/9291
Thrombophlebitis (Vascular disorders) | 2/9333 | 3/9291
Venous Thrombosis (Vascular disorders) | 2/9333 | 3/9291
Aortic Aneurysm Rupture (Vascular disorders) | 2/9333 | 1/9291
Arterial Occlusive Disease (Vascular disorders) | 2/9333 | 2/9291
Arteriosclerosis Obliterans (Vascular disorders) | 1/9333 | 2/9291
Arteriovenous Fistula (Vascular disorders) | 2/9333 | 1/9291
Artery Dissection (Vascular disorders) | 2/9333 | 0/9291
Cardiovascular Insufficiency (Vascular disorders) | 2/9333 | 1/9291
Femoral Artery Occlusion (Vascular disorders) | 2/9333 | 2/9291
Iliac Artery Stenosis (Vascular disorders) | 1/9333 | 2/9291
Leriche Syndrome (Vascular disorders) | 2/9333 | 1/9291
Shock Haemorrhagic (Vascular disorders) | 2/9333 | 0/9291
Thrombophlebitis Superficial (Vascular disorders) | 2/9333 | 1/9291
Thrombosis (Vascular disorders) | 2/9333 | 0/9291
Venous Thrombosis Limb (Vascular disorders) | 0/9333 | 2/9291
Aneurysm (Vascular disorders) | 0/9333 | 1/9291
Aneurysm Ruptured (Vascular disorders) | 1/9333 | 0/9291
Angiodysplasia (Vascular disorders) | 1/9333 | 0/9291
Aortic Dilatation (Vascular disorders) | 1/9333 | 1/9291
Arterial Disorder (Vascular disorders) | 1/9333 | 0/9291
Arterial Rupture (Vascular disorders) | 0/9333 | 1/9291
Arteritis (Vascular disorders) | 0/9333 | 1/9291
Bleeding Varicose Vein (Vascular disorders) | 1/9333 | 0/9291
Blood Pressure Inadequately Controlled (Vascular disorders) | 0/9333 | 1/9291
Embolism (Vascular disorders) | 1/9333 | 0/9291
Embolism Venous (Vascular disorders) | 1/9333 | 0/9291
Extremity Necrosis (Vascular disorders) | 1/9333 | 1/9291
Femoral Arterial Stenosis (Vascular disorders) | 0/9333 | 1/9291
Haemodynamic Instability (Vascular disorders) | 1/9333 | 0/9291
Iliac Artery Occlusion (Vascular disorders) | 0/9333 | 1/9291
Iliac Artery Thrombosis (Vascular disorders) | 1/9333 | 0/9291
Peripheral Artery Aneurysm (Vascular disorders) | 0/9333 | 1/9291
Peripheral Artery Dissection (Vascular disorders) | 1/9333 | 0/9291
Peripheral Embolism (Vascular disorders) | 1/9333 | 1/9291
Phlebitis (Vascular disorders) | 0/9333 | 1/9291
Reperfusion Injury (Vascular disorders) | 0/9333 | 1/9291
Subclavian Artery Stenosis (Vascular disorders) | 0/9333 | 1/9291
Subclavian Artery Thrombosis (Vascular disorders) | 0/9333 | 1/9291
Subclavian Vein Thrombosis (Vascular disorders) | 1/9333 | 0/9291
Vascular Occlusion (Vascular disorders) | 1/9333 | 0/9291
Vasculitis (Vascular disorders) | 1/9333 | 0/9291
Vena Cava Thrombosis (Vascular disorders) | 1/9333 | 0/9291
Venous Insufficiency (Vascular disorders) | 0/9333 | 1/9291
Wound Haemorrhage (Skin and subcutaneous tissue disorders) | 1/9333 | 0/9291
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | TICAGRELOR | CLOPIDOGREL
Headache (Nervous system disorders) | 621/9333 | 565/9291
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1106/9333 | 623/9291
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 566/9333 | 317/9291
Cough (Respiratory, thoracic and mediastinal disorders) | 490/9333 | 467/9291

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
An Investigator agrees to provide a copy of the publication to AstraZeneca (AZ) for review at least 60 days in advance of submission for publication. Investigators in multicenter (MC) studies agree to postpone MC publications until the earlier of the date of the first AZ-authorized MC publication or a period up to 18 months from study completion at all sites.